| 1 | The International Diabetes Closed Loop (iDCL) trial |
|---|-----------------------------------------------------|
| 2 | Clinical Acceptance of the Artificial Pancreas in |
| 2 | Padiatrics |

A Study of t:slim X2 with Control-IQ Technology

| 5 | <u>Study Sponsor</u> |
|------------|--------------------------------------------------------|
| 6 | Marc Breton |
| 7 | University of Virginia |
| 8 | Center for Diabetes Technology |
| 9 | Protocol Chair |
| 10 | R. Paul Wadwa, MD |
| 11 | Barbara Davis Center |
| 12 | University of Colorado |
| 13 | Participating Institutions |
| 14 | University of Virginia, Charlottesville, Virginia |
| 15 | Barbara Davis Center, University of Colorado, Colorado |
| 16 | Stanford University, California |
| 17 | Yale University, Connecticut |
| 18 | <b>Coordinating Center</b> |
| 19 | Jaeb Center for Health Research |
| 20 | |
| 21 | |
| <i>L</i> 1 | |
| 22 | |
| 23 | Version Number: v2.5 |
| 24 | May 24, 2019 |
| ∠+ | 141ay 27, 2017 |

| Sponsor Chair / IDE Chair | |
|---|---|
| Name, degree | Marc Breton |
| Institution Name | University of Virginia, Center for Diabetes Technology |
| Protocol Chair/Director | |
| Name, degree | R. Paul Wadwa, MD |
| Institution Name | Barbara Davis Center, University of Colorado |
| JCHR Coordinating Center Director | |
| Name, degree | Katrina Ruedy, MSPH |
| Institution Name | Jaeb Center for Health Research |
| Medical Monitor | |
| Name, degree | Roy Beck, M.D., Ph.D. |
| Institution Name | Jaeb Center for Health Research |

| Version<br>Number | Author(s) | Approver | Effective<br>Date | Revision Description |
|---|---|---|---|---|
| 1.0 | R. Paul Wadwa | R. Paul Wadwa | 15NOV2018 | Original protocol. |
| | Daniel Cherñavvsky | | | |
| | Katrina Ruedy | | | |
| | Roy Beck | | | |
| 1.1 | Jessica Rusnak | Daniel<br>Cherñavvsky | 21NOV2018 | |
| 1.2 | Sarah Borgman | Katrina Ruedy | 28NOV2018 | |
| 2.0 | Mary Oliveri | Daniel<br>Cherñavvsky | 10DEC2018 | Modified study design to include extension phase to the experimental group |
| 2.1 | Katrina Ruedy | Daniel<br>Cherñavvsky | 20Dec2018 | Clarifications added for consistency throughout protocol |
| 2.2 | Jessica Rusnak | Daniel<br>Cherñavvsky | 15Jan2019 | Adding inclusion criteria and clarification regarding use of Basal IQ feature; updated incorrect section references |
| 2.3 | Jessica Rusnak | Katrina Ruedy | 4Feb2019 | Removing and adding questionnaires to be completed by participants and parents/guardians |
| 2.4 | Katrina Ruedy | Daniel<br>Cherñavvsky | 01Apr2019 | Correcting discrepancies in revised questionnaire descriptions and other minor clarifications. |
| 2.5 | Katrina Ruedy | Marc Breton | 01Jun2019 | Corrections to statistical analysis chapter; update of Sponsor name from Daniel Cherñavvsky to Marc Breton |

| 31 | CHAPTER 1: BACKGROUND INFORMATION | 19 |
|----|----------------------------------------------------------------|----|
| 32 | 1.1 Introduction. | 19 |
| 33 | 1.2 Rationale | 22 |
| 34 | 1.3 Potential Risks and Benefits of the Investigational Device | 22 |
| 35 | 1.3.1 Known Potential Risks | 22 |
| 36 | 1.3.1.1 Venipuncture Risks | 22 |
| 37 | 1.3.1.2 Fingerstick Risks | 22 |
| 38 | 1.3.1.3 Subcutaneous Catheter Risks (CGM) | 22 |
| 39 | 1.3.1.4 Risk of Hypoglycemia | 23 |
| 40 | 1.3.1.5 Risk of Hyperglycemia | 23 |
| 41 | 1.3.1.6 Risk of Device Reuse | 23 |
| 42 | 1.3.1.7 Questionnaire | 24 |
| 43 | 1.3.1.8 Other Risks | 24 |
| 44 | 1.3.2 Known Potential Benefits | 24 |
| 45 | 1.3.3 Risk Assessment | 24 |
| 46 | 1.4 General Considerations | 25 |
| 47 | CHAPTER 2: STUDY ENROLLMENT AND SCREENING | 26 |
| 48 | 2.1 Participant Recruitment and Enrollment | 26 |
| 49 | 2.1.1 Informed Consent and Authorization Procedures | 26 |
| 50 | 2.2 Participant Inclusion Criteria | 27 |
| 51 | 2.3 Participant Exclusion Criteria | 28 |
| 52 | 2.4 Screening Procedures | 28 |
| 53 | 2.4.1 Data Collection and Testing | 28 |
| 54 | CHAPTER 3: RUN-IN PHASE | 30 |
| 55 | 3.1 Run-in Phase Overview | 30 |
| 56 | 3.2 Initiation of CGM | 30 |
| 57 | 3.3 Initiation of Pump | 30 |
| 58 | 3.4 Blood Glucose and Ketone Testing | 31 |
| 59 | 3.5 Assessment of Successful Completion of the Run-in Phase | 32 |
| 60 | 3.6 Optimization of Insulin Pump Settings | 33 |
| 61 | CHAPTER 4: RANDOMIZATION VISIT | 34 |

| 62 | 4.1 Randomization Visit | 34 |
|----|--------------------------------------------------------------------|----|
| 63 | 4.1.1 HbA1c | 34 |
| 64 | 4.1.2 Baseline C-Peptide Assessment | 34 |
| 65 | 4.1.3 Randomization | 34 |
| 66 | 4.1.4 Questionnaires | 35 |
| 67 | CHAPTER 5: MAIN STUDY PROCEDURES | |
| 68 | 5.1 Procedures for the CLC Group | |
| 69 | 5.2 Study System Training | 36 |
| 70 | 5.2.1 System Initiation | |
| 71 | 5.2.2 Home Use of the Study System | |
| 72 | 5.2.3 Study Device Download | 38 |
| 73 | 5.2.4 1-Week Phone Contact | 38 |
| 74 | 5.2.5 2-Week Visit (Training Review and Insulin Pump Optimization) | 38 |
| 75 | 5.3 Procedures for the SC Group | 39 |
| 76 | 5.3.1 Study Device Data Download | 39 |
| 77 | 5.3.2 1-Week Phone Contact | 39 |
| 78 | 5.3.3 2-Week Visit (Training Review and Insulin Pump Optimization) | 39 |
| 79 | 5.4 Follow-up Visits and Phone Contacts for Both Groups | 40 |
| 80 | 5.4.1 Follow-up Visits | 40 |
| 81 | 5.4.1.1 Procedures at Follow-up Visits | 40 |
| 82 | 5.4.2 Phone Contacts | 40 |
| 83 | 5.4.3 Data from Study Devices | 41 |
| 84 | 5.4.4 16-Week Final First Phase Visit | 41 |
| 85 | 5.5 Early Termination Visit (If Applicable) | 41 |
| 86 | 5.6 Unscheduled Visits | 41 |
| 87 | 5.7 Participant Access to Study Device at Study Closure | 41 |
| 88 | CHAPTER 6: EXTENSION PHASE PROCEDURES | 42 |
| 89 | 6.1 Closed Loop Control Participants | 42 |
| 90 | 6.2 SC Group Participants | 42 |
| 91 | 6.3 Early Termination Visit (If Applicable) | 43 |
| 92 | 6.4 Unscheduled Visits | 43 |
| 93 | 6.5 Participant Access to Study Device at Study Closure | 43 |

| 94 | CHAPTER 7: STUDY DEVICES | 44 |
|---|---|---|
| 95 | 7.1 Description of the Investigational Device | 44 |
| 96 | 7.1.1 Insulin Pump | 44 |
| 97 | 7.1.2 Continuous Glucose Monitoring | 44 |
| 98 | 7.1.3 Blood Glucose Meter and Strips | 44 |
| 99 | 7.1.4 Ketone Meter and Strips | 44 |
| 100 | 7.1.5 Study Device Accountability Procedures | 44 |
| 101 | 7.1.6 Blood Ketone Testing | 44 |
| 102 | 7.2 Safety Measures | 44 |
| 103 | 7.2.1 CGM Calibration | 44 |
| 104 | 7.2.2 System Failure | 45 |
| 105 | 7.2.3 Hypoglycemia Threshold Alert and Safety Protocol | 45 |
| 106 | 7.2.4 Hyperglycemia Threshold Alert and Safety Protocol | 45 |
| 107 | CHAPTER 8: TESTING PROCEDURES AND QUESTIONNAIRES | 47 |
| 108 | 8.1 Laboratory Testing | 47 |
| 109 | 8.1.1 Comprehensive Metabolic Panel (CMP) | 47 |
| 110 | 8.1.2 HbA1c: | 47 |
| 111 | 8.1.3 Urine Pregnancy: | 47 |
| 112 | 8.1.4 C-peptide and Glucose | |
| 113 | 8.2 Questionnaires | 47 |
| 114 | 8.2.1 Clarke's Hypoglycemia Awareness Scale – Child and Parent | 48 |
| 115 | 8.2.2 Hypoglycemia Fear Survey (HFS-II)/Low Blood Sugar Survey – | |
| 116 | Child and Parent | |
| 117 | 8.2.3 Problem Areas In Diabetes Survey (PAID) – Child and Parent | 48 |
| 118 | 8.2.4 PedsQL Diabetes Module – Child and Parent | |
| 119 | 8.2.5 INSPIRE Survey – Child and Parent | 49 |
| 120 | 8.2.6 Pittsburgh Sleep Quality Index (PSQI) – Parent | |
| 121 | 8.2.7 System Usability Scale (SUS) – Closed-Loop participants only | 49 |
| 122 | CHAPTER 9: ADVERSE EVENTS, DEVICE ISSUES, AND STOPPING RULES | |
| 123 | 9.1 Adverse Events | |
| 124 | 9.1.1 Definitions | |
| 125 | 9.1.2 Reportable Adverse Events | 51 |
| 126 | 9.1.2.1 Hypoglycemic Events | 51 |

| 127 | 9.1.2.2 Hyperglycemic Events/Diabetic Ketoacidosis | 51 |
|---|---|---|
| 128 | 9.1.3 Relationship of Adverse Event to Study Device | 52 |
| 129 | 9.1.4 Intensity of Adverse Event | 52 |
| 130 | 9.1.5 Coding of Adverse Events | 53 |
| 131 | 9.1.6 Outcome of Adverse Event | 53 |
| 132 | 9.2 Reportable Device Issues | 54 |
| 133 | 9.3 Pregnancy Reporting | 54 |
| 134 | 9.4 Timing of Event Reporting | 54 |
| 135 | 9.5 Stopping Criteria | 55 |
| 136 | 9.5.1 Participant Discontinuation of Study Device | 55 |
| 137 | 9.5.2 Criteria for Suspending or Stopping Overall Study | 55 |
| 138 | 9.6 Independent Safety Oversight | 55 |
| 139 | 9.7 Risks | 56 |
| 140 | CHAPTER 10: MISCELLANEOUS CONSIDERATIONS | 57 |
| 141 | 10.1 Drugs Used as Part of the Protocol | 57 |
| 142 | 10.2 Prohibited Medications, Treatments, and Procedures | 57 |
| 143 | 10.3 Participant Withdrawal | 57 |
| 144 | 10.4 Confidentiality | 57 |
| 145 | CHAPTER 11: STATISTICAL CONSIDERATION | 58 |
| 146 | 11.1 Statistical and Analytical Plans | 58 |
| 147 | 11.2 Statistical Hypotheses | 58 |
| 148 | 11.3 Sample Size | 58 |
| 149 | 11.4 Outcome Measures | 59 |
| 150 | 11.4.1 Primary Efficacy Endpoint | 59 |
| 151 | 11.4.2 Secondary Efficacy Endpoints | 59 |
| 152 | 11.4.2.1 Secondary Efficacy Endpoints Included in Hierarchical Analysis | 59 |
| 153 | 11.4.2.2 Other Secondary Efficacy Endpoints | 59 |
| 154 | 11.4.2.3 Safety Analyses | t defined. |
| 155 | 11.4.3 CGM Metrics Calculations | 60 |
| 156 | 11.5 Analysis Datasets and Sensitivity Analyses | 61 |
| 157 | 11.5.1 Per Protocol Analyses | 61 |
| 158 | 11.5.2 Other Sensitivity Analyses | 61 |
| 159 | 11.6 Analysis of the Primary Efficacy Endpoint | 62 |

| 160 | 11.7 Analysis of the Secondary Endpoints | 62 |
|-----|-----------------------------------------------------|----|
| 161 | 11.7.1 Hierarchical Analyses | 62 |
| 162 | 11.7.2 Other Endpoint Analyses | 63 |
| 163 | 11.8 Safety Analyses | 64 |
| 164 | 11.9 Intervention Adherence | 65 |
| 165 | 11.10 Adherence and Retention Analyses | 66 |
| 166 | 11.11 Baseline Descriptive Statistics | 66 |
| 167 | 11.12 Device Issues | 66 |
| 168 | 11.13 Planned Interim Analyses | 67 |
| 169 | 11.14 Subgroup Analyses | 67 |
| 170 | 11.15 Multiple Comparison/Multiplicity | 68 |
| 171 | 11.16 Exploratory Analyses | 68 |
| 172 | CHAPTER 12: DATA COLLECTION AND MONITORING | 69 |
| 173 | 12.1 Case Report Forms and Device Data | 69 |
| 174 | 12.2 Study Records Retention | 69 |
| 175 | 12.3 Quality Assurance and Monitoring | 69 |
| 176 | 12.4 Protocol Deviations | 70 |
| 177 | CHAPTER 13: ETHICS/PROTECTION OF HUMAN PARTICIPANTS | |
| 178 | 13.1 Ethical Standard | 71 |
| 179 | 13.2 Institutional Review Boards | 71 |
| 180 | 13.3 Informed Consent Process | 71 |
| 181 | 13.3.1 Consent Procedures and Documentation | 71 |
| 182 | 13.3.2 Participant and Data Confidentiality | 71 |
| 100 | | |
| 183 | CHAPTER 14: REFERENCES | 73 |

# **LIST OF ABBREVIATIONS**

| ABBREVIATION | DEFINITION |
|--------------|-------------------------------------------|
| AP | Artificial Pancreas |
| BG | Blood Glucose |
| BT/BTLE | Bluetooth, Bluetooth low energy |
| CRF | Case Report Form |
| CGM | Continuous Glucose Monitoring System |
| CLC | Closed-Loop Control |
| CSII | Continuous Subcutaneous Insulin Injection |
| CTR | Control-to-Range |
| DiAs | Diabetes Assistant |
| DKA | Diabetic Ketoacidosis |
| EC | European Commission |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| HbA1c | Hemoglobin A1c |
| ID | Identification |
| iDCL | International Diabetes Closed Loop |
| IDE | Investigational Device Exemption |
| IOB | Insulin-on-Board |
| IQR | Interquartile Range |
| JDRF | Juvenile Diabetes Research Foundation |
| LGS | Low Glucose Suspend |
| PLGS | Predictive Low Glucose Suspend |
| POC | Point-of-Care |
| QA | Quality Assurance |
| QC | Quality Control |
| RBM | Risk-Based Monitoring |
| RCT | Randomized Control Trial |
| SC | Standard of Care group |
| SD | Standard Deviation |
| TDD | Total Daily Dose |
| UI | User Interface |

186

# Signature Page

The International Diabetes Closed Loop (iDCL) trial:
Clinical Acceptance of the Artificial Pancreas in Pediatrics
A Study of t:slim X2 with Control-IQ Technology

**Protocol Identifying Number: DCLP5 Pediatrics** 

IND/IDE Sponsor: University of Virginia

Version Number: v.2.5

195 **24MAY2019** 

188

192

193

| Protocol Chair | |
|---|---|
| Name, Institution | R. Paul Wadwa, M.D./ University of Colorado – Barbara Davis Center |
| Signature/Date | |
| Sponsor (IDE Holder) | |
| Name/Institution | Marc Breton/ University of Virginia |
| Signature/Date | |
| <b>Coordinating Center Director</b> | |
| Name, Institution | Katrina J. Ruedy, MSPH; Jaeb Center for Health Research |
| Signature/Date | |
| Medical Monitor | |
| Name, Institution | Roy Beck, MD, PhD; Jaeb Center for Health Research |
| Signature/Date | |

| 196 | CLINICAL CENTER PRINCIPAL INVESTIGATOR | OR ST. | ATEN | <b>IENT</b> | OF | |
|---|---|---|---|---|---|---|
| 197 | COMPLIANCE | | | | | |
| 198<br>199 | Protocol Title: The International Diabetes Closed Loop (iDCL) the Artificial Pancreas in Pediatrics- A Study of t:slim X2 with | | | | | of |
| 200 | Protocol Version/Date: v2.5 / 24MAY2019 | | | | | |
| 201<br>202<br>203<br>204<br>205<br>206 | I have read the protocol specified above. In my formal capacity as Investigator, my duties include ensuring the safety of the study part supervision and providing the Jaeb Center for Health Research, wit information, as outlined in the protocol. It is understood that all int study will be held strictly confidential and that this confidentiality is study staff at this clinical center. | icipants<br>h comp<br>formatio | s enrol<br>lete an<br>on pert | led undend timely aining t | er my y to the | |
| 207<br>208<br>209<br>210 | This trial will be carried out in accordance with ICH E6 Good Clinical Practice (GCP) and as required by the following: United States (US) Code of Federal Regulations (CFR) applicable to clinical studies (45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, 21 CFR Part 312, and/or 21 CFR Part 812). | | | | | |
| 211<br>212<br>213<br>214 | As the Principal Investigator, I will assure that no deviation from, of will take place without prior agreement from the sponsor and document institutional Review Board (IRB), or other approved Ethics Committo eliminate an immediate hazard(s) to the trial participants. | nented | approv | al from | the | у |
| 215<br>216<br>217<br>218 | All key personnel (all individuals responsible for the design and co<br>completed Human Participants Protection Training and Good Clini<br>Further, I agree to ensure that all staff members involved in the con<br>informed about their obligations in meeting the above commitment | cal Prac<br>duct of | ctice T | raining. | | |
| 219<br>220 | Investigator's Signature | Date: | dd | / | _ / | уу |
| 221 | Investigator's Name: | | | | | |
| 222 | Clinical Center Name/Number | | | | | |

# PROTOCOL SUMMARY

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| Title | The International Diabetes Closed Loop (iDCL) trial: Clinical Acceptance of the Artificial Pancreas in Pediatrics- A study of t:slim X2 with Control-IQ Technology |
| Précis | A randomized controlled trial of at-home closed loop system vs. standard of care (defined as either sensor-augmented pump or any kind of low predictive low blood glucose suspend [PLGS; LGS] if participant is currently using) in youth age 6 to 13 years old. |
| Investigational Device | t:slim X2 with Control-IQ and Dexcom G6 system |
| Objectives | The objective of the study is to assess efficacy and safety of a closed loop control (CLC) system (t:slim X2 with Control-IQ Technology) in a randomized controlled trial with partial crossover. |
| Study Design | First phase a 16-week parallel group randomized clinical trial with 3:1 randomization to intervention with the closed loop system vs. standard of care (SC); followed by a 12-week period where the Standard of Care (SC) group will transition to use CLC and the experimental arm will extend the use of CLC for the same period |
| Number of Clinical Centers | Up to 4 US clinical centers |
| Endpoint | The primary outcome for the first phase is time in target range 70-180 mg/dL measured by CGM in CLC group vs. SC group over 16 weeks |
| | The primary outcome for the extension phase is improving time in range 70-180 mg/dL by CGM when SC (control group) transitions to t:slim X2 with Control-IQ compared with the same group during the Main Phase. |
| Population | <ul> <li>Key Inclusion Criteria</li> <li>Type 1 Diabetes</li> <li>Ages ≥ 6 and ≤ 13 years old</li> <li>Key Exclusion Criteria</li> <li>Use of any non-insulin glucose-lowering agents except metformin</li> <li>Actively using any other closed-loop system</li> </ul> |
| Sample Size | First phase: Up to 150 screened participants with the goal of randomizing 100 participants in this 16-week randomized trial. Extension phase will consist of a partial crossover: All randomized participants will participate in an extension phase for another 12 weeks (total 28 weeks). The SC group (control group) will crossover to use Tandem t:slim X2 with Control-IQ for 12 weeks. The experimental arm will continue on the Control-IQ for 12 weeks. |
| Treatment Groups | <ul> <li>Intervention Group: t:slim X2 with Control-IQ Technology and Study CGM.</li> <li>Control Group: Standard of care (SC) (defined as either sensor-augmented pump or any kind of low or predictive low blood glucose suspend [PLGS; LGS] if participant is currently using), and study CGM</li> <li>All participants will be offered to extend the study for 12 weeks and the SC group will use the t:slim X2 with Control-IQ System after the first 16-week phase</li> </ul> |
| Participant Duration | 16-20 weeks (depending on duration of run-in phase) plus ~12-week extension phase |

| PARTICIPANT AREA | DESCRIPTION |
|---|---|
| Protocol Overview/Synopsis | After consent is signed, eligibility will be assessed. Eligible participants not currently using an insulin pump and Dexcom G4, G5 or Dexcom G6 CGM with minimum data requirements will initiate a run-in phase of 2 to 4 weeks that will be customized based on whether the participant is already a pump or CGM user. Participants who skip or successfully complete the run-in will be randomly assigned 3:1 to the use of closed-loop control (CLC group) system using Tandem t:slim X2 with Control-IQ Technology vs SC for 16 weeks. All participants will be provided the option of using t:slim X2 with Control-IQ system in a 12 week Extension Phase. [Figure 1] |



226

Figure 1: Study Design: Participants Randomized 3:1 Control-IQ Control (CLC) vs. Standard of Care (SC) Groups. Extension phase with partial crossover of SC group switching to use Control IQ.

## **SCHEMATIC OF STUDY DESIGN**

### **Screening/Enrollment Visit**

- Eligibility assessment and informed consent
- HbA1c from local lab or POC device and central lab sample
- Device download and adherence assessment for current CGM user



<sup>\*</sup>Current use of insulin pump and Dexcom G4, G5, or G6 CGM with readings captured on at least 11 out of the previous 14 days

Figure 2: Schematic of Complete Study Design

230231



Figure 3: Schematic of Study Design (Post-Randomization)

| | Pre | Pre | 0 | 1w | 2w | 4w | 6w | 8w | 10w | 12w | 14w | 16w |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit (V) or Phone (P) | V | V | V | P | V | P | P | V | P | P | P | V |
| Comment | Screen/<br>Enroll | Run-in | Rand | | | | | | | | | |
| Eligibility Assessment | X | X | X | | | | | | | | | |
| HbA1c (DCA Vantage or similar point of care device, or local lab) | X | | X | | | | | | | | | X |
| HbA1c (Central lab) | | | X | | | | | | | | | X |
| C-peptide (Central lab) and blood glucose assessment | | | X | | | | | | | | | |
| Pregnancy test (females of child-bearing potential) | X | | X | | | | | X | | | | X |
| Device Data download(s) | X | X | X | X | X | X | X | X | X | X | X | X |
| Review diabetes management and AEs | | X | X | X | X | X | X | X | X | | | X |
| Questionnaires as defined in section 8.2 | | | X | | | | | | | | | X |

**Table 1. Schedule of Study Visits and Procedures (Primary Study Phase)** 

| Experimental Group | 20w | 24w | 28w |
|---|---|---|---|
| Visit (V) or Phone (P) | P | P | V |
| Comment | | | |
| Eligibility Assessment | | | |
| HbA1c (DCA Vantage or similar point of care device, or local lab) | | | X |
| HbA1c (Central lab) | | | X |
| C-peptide (Central lab) and blood glucose assessment | | | |
| Pregnancy test (females of child-bearing potential) | | | X |
| Device Data download(s) | X | X | X |
| Review diabetes management and AEs | X | X | X |
| Questionnaires as defined in section 8.2 | | | X |

Table 2: Schedule of Visits and Procedures (Extension Phase for Experimental Group)

| 249 |
|-----|
| 250 |
| 251 |
| 252 |
| 253 |
| 254 |
| 255 |
| 256 |
| 257 |
| 258 |
| 259 |

| Control Group | 17w | 19w | 21w | 23w | 25w | 28w |
|---|---|---|---|---|---|---|
| Visit (V) or Phone (P) | P | P | P | V | P | V |
| Comment | | | | | | |
| Eligibility Assessment | | | | | | |
| HbA1c (DCA Vantage or similar point of care device, or local lab) | | | | | | X |
| HbA1c (Central lab) | | | | | | X |
| C-peptide (Central lab) and blood glucose assessment | | | | | | |
| Pregnancy test (females of child-bearing potential) | | | | X | | X |
| Device Data download(s) | X | X | X | X | X | X |
| Review diabetes management and AEs | X | X | X | X | X | X |
| Questionnaires as defined in section 8.2 | | | | | | X |

**Table 3: Schedule of Visits and Procedures (Extension Phase for SC Group)** 

260

261

#### 1.1 Introduction

- The Tandem X2 insulin pump with Control-IQ Technology is a third-generation closed-loop
- 267 control (CLC) system retaining the same control algorithm that was initially tested by UVA's DiAs
- system and then implemented in the inControl system (TypeZero Technologies, Inc.). DiAs is
- described in 13 IDEs (see IDEs 1-12 and 14 in the list below) and inControl is described on the
- 270 rest of IDEs mentioned below (i.e.in IDEs G160097, G160181, G150240, G140169/S010). For
- complete algorithmic and clinical background, we refer to these IDEs and to a number of scientific
- 272 publications that describe glycemic control outcomes and clinical impressions from the use of
- these systems (see list of 25 peer-reviewed papers and scientific presentations under Bibliography).
- Overall, this control algorithm has been implemented in two mobile platforms (DiAs and
- inControl) and has been tested in 30 clinical trials by 450 adults and children with type 1 diabetes
- for over 350,000 hours of use to date in the U.S. and overseas.
- As described in the Background, this project is a result from a sequence of clinical trials that have
- 278 tested extensively the control system and in several centers in the U.S. and overseas. The following
- 279 21 IDEs reflect this progress:
- 1. IDE #G110095: Feasibility study of closed loop control in type 1 diabetes using heart rate monitoring as an exercise marker, approved 10/08/2011;
- 282 2. IDE #G120032: Early feasibility (pilot) study of outpatient control-to-range; 3/2/2012;
- 3. IDE #G120210: Early feasibility study 2 of outpatient control-to-range; 10/12/2012;
- 4. IDE #G130118: DiAs control-to-range nocturnal closed-loop camp study; 6/19/2013;
- 5. IDE #G130121: Optimizing closed-loop control of type 1 diabetes mellitus in adolescents; 6/19/2013;
- 6. IDE# G130142: Closed loop control in adolescents using heart rate as exercise indicator; 7/16/13;
- 7. IDE #G130143: Early feasibility study of adaptive advisory/automated (AAA) control of type 1 diabetes; 7/19/2013;
- 8. IDE #G140066: Full day and night closed-loop with DiAs platform; 5/9/14.
- 9. IDE #G140068: Unified Safety System (USS) Virginia Closed Loop versus sensor augmented pump therapy overnight in type 1 diabetes; 5/14/2014;
- 294 10. IDE #G140089: Outpatient control-to-range: Safety and efficacy with day-and-night in-home use; 6/6/2014;
- 11. IDE #G140169: Unified Safety System (USS) Virginia Closed-Loop versus Sensor
   Augmented Pump (SAP) therapy for hypoglycemia reduction in type 1 diabetes; 10/3/2014.
- 12. IDE #G150221: Reducing risks and improving glucose control during extended exercise in youth with T1DM: The AP Ski Camp; 11/09/2015;

- 13. IDE #G150240: Project Nightlight: Efficacy and system acceptance of dinner/night vs. 24 hr
   closed loop control; 11/12/2015;
- 302 14. IDE #G160047: Closed-loop in young children 5-8 years old using DiAs platform; 303 03/29/2016;
- 304 15. IDE #G160097: Clinical Acceptance of the Artificial Pancreas: the International Diabetes
   305 Closed-Loop (iDCL) Trial/Research Site Training Protocol; 06/03/16.
- 306 16. IDE#G160181: PROTOCOL 1 for "Clinical Acceptance of the Artificial Pancreas: The
   307 International Diabetes Closed Loop (iDCL) Trial; 09/21/16
- 308 17. IDE#G170255: Protocol 3 for "Pilot Trial of t:slim X2 with Control-IQ
   309 Technology";11/16/17 and IDE#G170255/S001 Protocol 3 for "Training Study of t:slim X2 with Control-IQ Technology"; 11/16/17
- 18. IDE#G170267: "Real-Time Monitoring and Glucose Control During Winter-Sport Exercise
   in Youth with Type 1 Diabetes: The AP Ski Camp Continued"; 11/21/17
- 19. IDE#G150240/S008: A long-term home use study, enrolling 18-70 years old TID
   participants since January 2018; it is anticipated that this study will be completed April 2019.
- 20. IDE#G170255: A pilot study of 5 adult subjects completed in December 2017.
- 21. IDE#G170267: Three 48-hour winter ski camps trial T1D participants; one site enrolled 13-
- 18 years old participants in January 2018. The other two sites enrolled participants aged 6-12
- years old. At the conclusion of these ski camps, subjects continued with the study device for
- 319 72 hours use at home (March & April 2018).
- 320 In the G170255 pilot study (mean age 52.8 yrs; 3F/2M, mean A1c 6.5%), the system was
- 321 challenged with a variety of scenarios including: Pump disconnection, CGM sensor removal
- 322 without stopping session, CGM sensor change, Basal Rate change, Cartridge Change, Extended
- 323 Bolus, Calibration at non-ideal conditions, Stopping Control-IQ, Reset Sleep Time, Restaurant
- 324 Meals and Exercise (treadmill/walk). The study demonstrated excellent connectivity with 98%
- time in closed-loop control and 94%-time CGM is available during 196 hours of use. [28]
- The results of the home portion of the IDE#G170267/ski camp trial (Table 5) were as follow: The
- 327 Control-IQ significantly improved time in target range 70-180 mg/dL (71.0±6.6 vs. 52.8±13.5%;
- 328 p=0.001) and mean sensor glucose (153.6 $\pm$ 13.5 vs. 180.2 $\pm$ 23.1 mg/dL; p=0.003) without
- 329 increasing hypoglycemia time <70 mg/dL (1.7 [1.3-2.1] vs. 0.9 [0.3-2.7]%; ns). The HCL system
- was active for 94.4% of the study period. Subjects reported that use of the system was associated
- with less time thinking about diabetes, decreased worry about blood sugars, and decreased burden
- in managing diabetes. [33]
- No AE or SAE happened during these trials related to the equipment used.

| METRIC (COMPUTED DURING CLOSED-LOOP USE) | OVERALL | DAYTIME | NIGHTTIME |
|------------------------------------------|---------|---------|-----------|
| Mean glucose (mg/dL) | 129 | 135 | 121 |
| Coefficient of variation (median) | 27% | 27% | 21% |
| % below 54 mg/dL (median) | 0.7% | 0.0% | 0.0% |
| % below 60 mg/dL (median) | 1.1% | 2.0% | 0.0% |
| % below 70 mg/dL (median) | 2.9% | 4.1% | 1.0% |
| Percent in range 70-180 mg/dL (mean) | 87% | 82% | 94% |
| % above 180 mg/dL (median) | 5% | 8% | 6% |
| % above 250 mg/dL (median) | 0% | 0% | 0% |
| % above 300 mg/dL (median) | 0% | 0% | 0% |

Table 4. Pilot Study results based on time in closed-loop

| | | OVERALL | | DAYTIN | ME [7AM - 11 P | NIGHTIME [11PM - 7AM] | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Control-<br>IQ | SAP | p-<br>value | Control-IQ | SAP | p-<br>value | Control-IQ | SAP | p-<br>value |
| 70 - 180 mg/dL<br>(%) | $71.0 \pm 6.6$ | $52.8 \pm 13.5$ | 0.001 | 69.1 ± 10.1 | 54.4 ± 14.2 | 0.010 | $74.9 \pm 10.1$ | $49.6 \pm 18.8$ | 0.001 |
| < 50 mg/dL (%) | 0 [0-0.1] | 0 [0-0.4] | ns | 0 [0-0] | 0 [0-0.6] | ns | 0 [0-0] | 0 [0-0] | ns |
| < 54 mg/dL (%) | 0.2 [0-0.5] | 0.2 [0-0.6] | ns | 0 [0-0.4] | 0.3 [0-0.9] | ns | 0 [0-0] | 0 [0-0] | ns |
| < 60 mg/dL (%) | 0.7 [0.2-1] | 0.5 [0-0.9] | ns | 0.3 [0-1.1] | 0.7 [0-1.3] | ns | 0 [0-0.2] | 0 [0-0] | ns |
| < 70 mg/dL (%) | 1.7 [1.3-<br>2.1] | 0.9 [0.3-2.7] | ns | 1.6 [0.7-2.6] | 1.4 [0.5-3.4] | ns | 0.7 [0-2.6] | 0 [0-0] | 0.190 |
| > 180 mg/dL (%) | $26.7 \pm 7.2$ | $44.7 \pm 13.8$ | 0.001 | $28.1 \pm 11.1$ | $42 \pm 14.4$ | 0.017 | $23.8 \pm 9.9$ | $49.9 \pm 19.3$ | 0.001 |
| > 250 mg/dL (%) | $7.2 \pm 4.5$ | $16.1 \pm 10.3$ | 0.015 | $8.3 \pm 6.4$ | $14.8 \pm 11$ | 0.097 | 5.2 ± 8 | $18.7 \pm 12.9$ | 0.007 |
| > 300 mg/dL (%) | $2.9 \pm 2.7$ | $5.3 \pm 3.9$ | 0.102 | $3.5 \pm 3.9$ | $4.4 \pm 4.5$ | ns | $1.8 \pm 4$ | $7.1 \pm 6.5$ | 0.030 |
| Mean glucose (mg/dL) | 153.6 ±<br>13.5 | $180.2 \pm 23.1$ | 0.003 | $157 \pm 20.2$ | $175.7 \pm 24.7$ | 0.064 | 147.1 ±<br>16.4 | 188.8 ± 30.2 | 0.001 |
| Coefficient of Variation (%) | $36.6 \pm 4.9$ | $36.5 \pm 5.4$ | ns | $35.7 \pm 5.3$ | $36.8 \pm 6.1$ | 0.185 | $33.4 \pm 7.1$ | $32.9 \pm 6.4$ | ns |
| Insulin use (U/day) | 33.2 ± 15.5 | $27.8 \pm 12.3$ | ns | $26.4 \pm 12.8$ | $22.3 \pm 9.6$ | ns | $6.8 \pm 2.8$ | 5.5 ± 3 | ns |
| CHO treatment (g) | 15.5 ± 16.9 | $35.5 \pm 55.5$ | ns | $14.7 \pm 16.7$ | $34.5 \pm 55.7$ | ns | $0.9 \pm 2$ | $1.2 \pm 2.6$ | ns |

### Table 5. Glycemic Outcomes Measured by CGM: Ski camp and home use trial

## **Closed-Loop Control System**

The Closed-Loop Control System contained in t-slim X2 with Control-IQ Technology is described in Master File MAF-2032/A008. Control-IQ Technology is derived from inControl previously described in IDE# G160097, G160181, G150240 and G140169/S010. The CLC is an "artificial pancreas" (AP) application that uses advanced closed loop control algorithms to automatically manage blood glucose levels for people with Type 1 Diabetes. The system modulates insulin to keep blood glucose in a targeted range. The system components include the t:slim X2 with Control-IQ Technology and the Dexcom CGM G6.



354

358

359

360

361

362363

364

365

366

367

368369

370

371

372

373

Figure 4. t:slim X2 with Control-IQ and Dexcom G6 system

#### **1.2 Rationale**

- 349 The objective of this randomized clinical trial is to assess the efficacy and safety of the Control-
- 350 IQ closed loop system over a 16-week period compared with standard of care. In addition, the data
- from this trial may be used for subsequent PMA application for this system.
- The 12-week extension phase will allow for additional exposure time to the Tandem t:slim X2 with Control-
- 353 IQ Technology and evaluation of the SC arm when crossover to use Control IQ for 12-week period.

## 1.3 Potential Risks and Benefits of the Investigational Device

- Risks and Benefits are detailed below. Loss of confidentiality is a potential risk; however, data are
- handled to minimize this risk. Hypoglycemia, hyperglycemia and ketone formation are always a
- risk in participants with type 1 diabetes and participants will be monitored for these events.

#### 1.3.1 Known Potential Risks

#### 1.3.1.1 Venipuncture Risks

A hollow needle/plastic tube will be placed in the arm for taking blood samples. Blood draws can cause some common reactions like pain, bruising, or redness at the sampling site. Less common reactions include bleeding from the sampling site, formation of a small blood clot or swelling of the vein and surrounding tissues, and fainting.

#### 1.3.1.2 Fingerstick Risks

About 1 drop of blood will be removed by fingerstick for measuring blood sugars and sometimes HbA1c or other tests. This is a standard method used to obtain blood for routine hospital laboratory tests. Pain is common at the time of lancing. In about 1 in 10 cases, a small amount of bleeding under the skin will produce a bruise. A small scar may persist for several weeks. The risk of local infection is less than 1 in 1000. This should not be a significant contributor to risks in this study as fingersticks are part of the usual care for people with diabetes.

#### 1.3.1.3 Subcutaneous Catheter Risks (CGM)

Participants using the CGM will be at low risk for developing a local skin infection at the site of the sensor needle placement. If a catheter is left under the skin for more than 24 hours, it is possible

- 374 to get an infection where it goes into the skin, with swelling, redness and pain. There may be
- 375 bleeding where the catheter is put in and bleeding under the skin causes a bruise (1 in 10 risk).
- 376 Study staff should verbally alert the participant that on rare occasions, the CGM may break and
- 377 leave a small portion of the sensor under the skin that may cause redness, swelling or pain at the
- 378 insertion site. The participant should be further instructed to notify the study coordinator
- 379 immediately if this occurs.

#### 1.3.1.4 Risk of Hypoglycemia

- 381 As with any person having type 1 diabetes and using insulin, there is always a risk of having a low
- 382 blood sugar (hypoglycemia). The frequency of hypoglycemia should be no more and possibly less
- 383 than it would be as part of daily living. Symptoms of hypoglycemia can include sweating,
- 384 jitteriness, and not feeling well. Just as at home, there is the possibility of fainting or seizures
- 385 (convulsions) and that for a few days the participant may not be as aware of symptoms of
- 386 hypoglycemia. A CGM functioning poorly and significantly over-reading glucose values could
- 387 lead to inappropriate insulin delivery.

## 1.3.1.5 Risk of Hyperglycemia

- 389 Hyperglycemia and ketonemia could occur if insulin delivery is attenuated or suspended for an
- 390 extended period or if the pump or infusion set is not working properly. A CGM functioning poorly
- 391 and significantly under-reading glucose values could lead to inappropriate suspension of insulin
- 392 delivery.

380

388

393

#### 1.3.1.6 Risk of Device Reuse

- 394 The study CGM system is labeled for single use only. The sensor (the component of the system
- 395 that enters the skin) will be single use only. The receiver, if used, is a hand-held device. The
- 396 transmitter and receiver may be reused during the study after cleaning the device using a hospital-
- 397 approved cleaning procedure. The transmitter is attached to the sensor but does not enter the skin.
- 398 Participants will be informed that FDA or relevant national authorities have approved these devices
- 399 for single use and that by using them among multiple patients, bloodborne pathogens (i.e. Hepatitis
- 400 B) may be spread through the use of multiple users.
- 401 The study insulin pump is labeled for single-patient use. During the study, this device may be
- 402 reused after cleaning adhering to a hospital-approved cleaning procedure. All infusion set
- 403 equipment will be single patient use only (infusion set insertion kits, tubing, cartridges etc.)
- 404 Participants will be informed that FDA or relevant national authorities typically approve the insulin
- 405 pump device for single use and that by using them among multiple patients, bloodborne pathogens
- 406 (i.e. Hepatitis B) may be spread through the use of multiple users.
- 407 The study blood glucose meter and blood ketone meter are labeled for single-patient use.
- 408 During the study, only one person can use each device as there are rare risks that bloodborne
- 409 pathogens (i.e. Hepatitis B) may be spread through the use of multiple users.

#### 410 **1.3.1.7 Questionnaire**

- 411 As part of the study, participants (parent and child) will complete questionnaires which include
- 412 questions about their private attitudes, feelings and behavior related to the investigational
- 413 equipment as well as managing diabetes. It is possible that some people may find these
- questionnaires to be mildly upsetting. Similar questionnaires have been used in previous research
- and these types of reactions have been uncommon.

#### 1.3.1.8 Other Risks

- Some participants may develop skin irritation or allergic reactions to the adhesives used to secure
- 418 the CGM, or to secure the insulin infusion sets for the continuous subcutaneous insulin infusion.
- 419 If these reactions occur, different adhesives or "under-taping" (such as with IV 3000, Tegaderm,
- 420 etc.) will be tried, sites will be rotated frequently, and a mild topical steroid cream or other
- 421 medication may be required.
- Whenever the skin is broken there is the possibility of an infection. The CGM and pump infusion
- sites are inserted under the skin. It is possible that any part that is inserted under the skin may
- 424 cause an infection. These occur very infrequently, but, if an infection was to occur, oral and/or
- 425 topical antibiotics can be used. The risk of skin problems could be greater if you use a sensor for
- longer than it is supposed to be used. Therefore, participants (and parents) will be carefully
- instructed about proper use of the sensor.
- Data downloaded from the CGM, pump, and the home glucose and ketone meter will be collected
- 429 for the study as measures of diabetes self-management behaviors. Some people
- may be uncomfortable with the researchers' having such detailed information about their daily
- diabetes habits.

432

439

416

#### 1.3.2 Known Potential Benefits

- One purpose of this research is to reduce the frequency of hypoglycemia and severe hypoglycemic
- events. Hypoglycemia is the number one fear of many individuals and families with someone who
- has type 1 diabetes and this fear often prevents optimal glycemic control.
- 436 It is expected that this protocol will yield increased knowledge about using an automated
- closed-loop system to control the glucose level and is intended to develop data to support a future
- 438 PMA-application. The individual participant may not benefit from study participation.

#### 1.3.3 Risk Assessment

- Based on the facts that (1) children and adolescents with diabetes experience mild hypoglycemia
- and hyperglycemia frequently as a consequence of the disease and its management, (2) the study
- intervention involves periodic automated insulin dosing that may reduce the likelihood of
- 443 hypoglycemia, and periodic automated attenuation of insulin delivery that may reduce the
- likelihood of hyperglycemia, (3) if any, hypo and/or hyperglycemia occur, mitigations are in place,
- and have been tested in prior studies using the investigational device system in the home setting,
- 446 that limit the likelihood of excessive insulin dosing or prolonged withdrawal of insulin, and (4)
- rapid reversal of hypoglycemia and hyperglycemia can be achieved, it is the assessment of the
- investigators that this protocol falls under DHHS 46.405 which is a minor increase over minimal

- risk. In addition, it is the belief of the investigators that this study also presents prospect of direct
- benefit to the participants and general benefit to others with diabetes.

### 451 **1.4 General Considerations**

- The study is being conducted in compliance with the policies described in the study policies
- document, with the ethical principles that have their origin in the Declaration of Helsinki, with the
- 454 protocol described herein, and with the standards of Good Clinical Practice (GCP).
- Whenever possible, data will be directly collected in electronic case report forms, which will be
- 456 considered the source data.
- There is no restriction on the number of participants to be enrolled by each clinical center toward
- 458 the overall recruitment goal.
- The protocol is considered a significant risk device study, due to the fact that the closed loop
- system is experimental. Therefore, an investigational device exemption (IDE) from the U.S. Food
- and Drug Administration (FDA) is required to conduct the study.

## **Chapter 2: Study Enrollment and Screening**

## 463 2.1 Participant Recruitment and Enrollment

462

- Enrollment will proceed with the goal of having 100 participants randomized for the first 16-week
- phase of this trial. A maximum of 150 individuals may be enrolled into screening for the study in
- order to achieve this goal considering an approximately 30% withdrawal and screen failure rate.
- For the extension phase, all 100 participants that were randomized and completed the main study
- will complete the 12-week extension phase. The participants randomized to SC in the main study
- will crossover to use t:slim x2 with Control IQ. The interventional arm in the main study will
- 470 continue using the Control IQ system for 12 additional weeks.
- 471 Study participants will be recruited from up to 4 clinical centers in the United States without regard
- 472 to gender, race, or ethnicity. There is no restriction on the number of participants to be enrolled
- by each clinical center toward the overall recruitment goal.
- The study team will make every effort to have the following minimum numbers of participants
- complete the trial in the specified subgroups at the time of enrollment:
- At least one-third of participants with HbA1c ≥8.0% and one-third of participants with HbA1c 477 <7.9%
- At least one-third of participants in the age range 6-10 and one-third of participants 11-13 years old
- At least 20% of participants who are on multiple daily injections (MDI) rather than pump
- At least 20% of participants who are CGM-naïve (defined as not using a CGM in the prior 3 months)

## 2.1.1 Informed Consent and Authorization Procedures

- Potential eligibility may be assessed as part of a routine-care examination. Before completing any
- procedures or collecting any data that are not part of usual care, written informed consent and child
- assent will be obtained.

- 487 A parent/legal guardian (referred to subsequently as "parent") will be provided with the Informed
- Consent Form to read and will be given the opportunity to ask questions. Potential participants
- 489 meeting the IRB's minimum age of assent will be given a Child Assent Form to read and discuss
- with his/her parents and study personnel. If the parent and child agree to participate, the Informed
- 491 Consent Form and Child Assent Form (if applicable) will be signed. A copy of the consent form
- will be provided to the participant and his/her parent and another copy will be added to the
- 493 participant's study record.
- 494 As part of the informed consent process, each participant and/or parent/legal guardian will be asked
- 495 to sign an authorization for release of personal information. The investigator, or his or her
- designee, will review the study-specific information that will be collected and to whom that

- 497 information will be disclosed. After speaking with the participant, questions will be answered
- about the details regarding authorization.
- 499 A participant is considered enrolled when the informed consent form and child assent (if
- applicable) has been signed.
- 501 **2.2 Participant Inclusion Criteria**
- Individuals must meet all of the following inclusion criteria in order to be eligible to participate in
- 503 the study.
- 1. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year
- and using insulin for at least 6 months
- 506 2. Familiarity and use of a carbohydrate ratio for meal boluses.
- 507 3. Age  $\geq$  6 and  $\leq$  13 years old
- 508 4. Weight  $\geq$ 25 kg and  $\leq$ 140 kg
- 5. For females, not currently known to be pregnant
- If female and sexually active, must agree to use a form of contraception to prevent pregnancy
- while a participant in the study. A negative serum or urine pregnancy test will be required for
- all females of child-bearing potential. Participants who become pregnant will be discontinued
- from the study. Also, participants who during the study develop and express the intention to
- become pregnant within the timespan of the study will be discontinued.
- 6. Living with one or more parent/legal guardian knowledgeable about emergency procedures for
- severe hypoglycemia and able to contact emergency services and study staff.
- 7. Willingness to suspend use of any personal closed loop system that they use at home for the
- duration of the clinical trial once the study CGM is in use
- 8. Investigator has confidence that the participant can successfully operate all study devices and
- is capable of adhering to the protocol
- 9. Willingness to switch to lispro (Humalog) or aspart (Novolog) if not using already, and to use
- no other insulin besides lispro (Humalog) or aspart (Novolog) during the study for participants
- using the t:slim X2. This includes:
- 524 o Participants randomized to Control IQ
- 525 o Participants on the SC group on MDI treatment that will be provided a Tandem
- 526 pump to switch to CSII
- 527 o Participates that are already in CSII randomized to SC during the extension phase
- 528 when transition to Control IQ
- 529 10. Total daily insulin dose (TDD) at least 10 U/day
- 530 11. Willingness not to start any new non-insulin glucose-lowering agent during the course of the
- trial (see section 2.3)

532 12. Participant and parent(s)/guardian(s) willingness to participate in all training sessions as directed by study staff.

## 534 **2.3 Participant Exclusion Criteria**

- Individuals meeting any of the following exclusion criteria at baseline will be excluded from study
- 536 participation.
- 1. Concurrent use of any non-insulin glucose-lowering agent other than metformin (including
- 538 GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas).
- 539 2. Hemophilia or any other bleeding disorder
- 3. A condition, which in the opinion of the investigator or designee, would put the participant or study at risk (specified on the study procedure manual)
- 542 4. Participation in another pharmaceutical or device trial at the time of enrollment or during the study
- 5. Employed by, or having immediate family members employed by Tandem Diabetes Care, Inc.,
- or having a direct supervisor at place of employment who is also directly involved in
- conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree
- relative who is directly involved in conducting the clinical trial

## 548 **2.4 Screening Procedures**

- After informed consent has been signed, a potential participant will be evaluated for study
- eligibility through the elicitation of a medical history, performance of a physical examination
- by study personnel and local laboratory testing if needed to screen for exclusionary medical
- 552 conditions.
- Individuals who do not initially meet study eligibility requirements may be rescreened at a later
- date per investigator discretion.

#### 555 **2.4.1 Data Collection and Testing**

- A standard physical exam (including vital signs and height and weight measurements) will be
- performed by the study investigator or designee (a physician, research physician, resident, fellow,
- nurse practitioner or a physician assistant).
- The following procedures will be performed/data collected/eligibility criteria checked and
- documented:
- Inclusion and exclusion criteria assessed
- Demographics (date of birth, sex, race and ethnicity)
- Contact information (retained at the clinical center and not entered into study database)
- Medical history
- Concomitant medications

- Physical examination to include:
- Weight, height
- Vital signs including measurement of blood pressure and pulse
- Comprehensive Metabolic Panel to assess kidney and liver functioning
- 570 Blood draw for:
- HbA1c level measured using the DCA Vantage or comparable point of care device or local lab
- 572 Measurement performed as part of usual clinical care prior to obtaining informed consent 573 for participation in the trial may be used
- o Measurement must be made within two weeks prior to enrollment
- 575 O Sample to be sent to a central lab
- Urine or serum pregnancy test for all women of child-bearing potential and sexually active.
- 577 Screening procedures will last approximately 1-2 hours.

611

612

#### 579 3.1 Run-in Phase Overview This phase may begin immediately after enrollment is complete or may be deferred for a maximum 580 581 of 28 days. The purpose of this run-in phase is to 1) assess compliance with study procedures, 2) 582 to introduce the study CGM to study participants without current use of a CGM and 3) to introduce 583 an insulin pump to participants who have not previously used an insulin pump. 584 Participants who currently use an insulin pump and a Dexcom G4, G5 or G6 with CGM data 585 captured on at least 11 out of the previous 14 days prior to the time of enrollment can skip the runin phase. If a participant is using a pump with a Low Glucose Suspend (LGS) feature, they will be 586 587 allowed to continue using this feature. Participants who do not currently use a Dexcom G4, G5, or 588 G6 CGM will be required to participate in the CGM run-in phase. Participants currently using a 589 Dexcom G4, G5, or G6 CGM with CGM readings captured on fewer than 11 out of the previous 590 14 days prior to time of enrollment will be required to participate in the CGM run-in phase. During the CGM run-in phase, participants will use the study CGM for a minimum of 11 days with a goal 591 592 of at least 14 days. 593 All participants and their parent(s) will receive training on the study CGM as detailed below. This 594 will be an unblinded use of the study CGM. 595 Additionally, MDI and study pump naïve participants will participate in a pump run-in phase that 596 will run 2 to 6 weeks before randomization is assigned. If both pump run-in phase and CGM run-597 in phase are indicated, they will run concurrently. Training is detailed below. 598 599 3.2 Initiation of CGM 600 The participant will be provided with sensors and instructed to use the study CGM on a daily basis. 601 Training will be provided to participants not experienced with CGM use as to how to use the CGM 602 in real-time to make management decisions and how to review the data after an upload for 603 retrospective review. Participants using a personal CGM prior to the study will discontinue the 604 personal CGM beginning in this period. 605 The participant will be observed placing the sensor. The study CGM user's guide will be provided 606 for the participant to take home. 607 3.3 Initiation of Pump 608 Pump-naïve participants will use the study insulin pump and CGM for up to 4 weeks before 609 randomization is assigned.

Participants who are pump-naïve will be provided with a study pump similar to the pump used

with the closed-loop system, but with the closed-loop control feature either absent or deactivated

and will be instructed to use the pump on a daily basis. An initial basal insulin profile will be

- customized on a per-participant basis. Total daily insulin dose will be reduced by approximately
- 614 20% as a general rule, with a recommended method outlined in a separate procedures' manual.
- Further adjustments to total daily dose (TDD) and intraday basal rate profile may be made during
- the course of the run-in period that can be concomitant with the CGM run-in phase.
- Participants and parent(s) will complete training on the study pump as detailed below.
- The participant will be fully instructed on the study insulin pump. A qualified system trainer will conduct the training and in particular discuss differences from their home pump in important aspects such as calculation of insulin on board (IOB) and correction boluses.
- The study pump will have the Basal-IQ feature, and participants will be able to use this feature at investigator discretion.
- Additional topics are not limited to but may include: infusion site initiation, cartridge/priming
- procedures, setting up the pump, charging the pump, navigation through menus, bolus
- procedures including stopping a bolus, etc.
- For pump-naïve participants, the study team will assist the participant in study pump infusion site initiation and will start the participant on the study pump. The study pump will be programmed with the participant's insulin requirements.
- The participant will be supervised with the study pump during at least one meal or snack bolus to ensure participant understanding of the pump features.
- The participant will be encouraged to review the literature provided with the pump and infusion sets after the training is completed.
- Note: For the extension phase, participants in the control group will be trained on the use of the Control IO system. Follow up phone contacts and in-clinic visits are described in Table 3.

## 3.4 Blood Glucose and Ketone Testing

- Participants will receive supplies for blood glucose and ketone testing.
- Blood glucose testing

633

636

- 640 Participants will be provided with a study blood glucose meter, test strips, and standard control solution to perform quality control (QC) testing at home per manufacturer guidelines.
- 642 O All study blood glucose meters will be QC tested with control solution if available during 643 all office visits. A tested meter will not be used in a study if it does not read within the target 644 range at each concentration per manufacturer labeling. The participant will be instructed to 645 contact study staff for a replacement of the meter, test strips, and control solution if a meter 646 fails QC testing at home.

- 647 O Participants will be reminded to use the study blood glucose meter for all fingerstick BGs during the study.
- o Participants will be given guidelines for treatment of low or high blood glucose.
- Blood ketone testing
- 651 O Participants will be provided with a study blood ketone meter, test strips, and standard control solution to perform QC testing at home per manufacturer guidelines.
- 653 O All study blood ketone meters will be QC tested with control solution if available during 654 all office visits. A tested meter will not be used in a study if it does not read within the target 655 range at each concentration per manufacturer labeling. The participant will be instructed to 656 contact study staff for a replacement of the meter, test strips, and control solution if a meter 657 fails QC testing at home.
- o Participants will be instructed to perform blood ketone testing as described in section 7.1.6.
- o Participants will be given guidelines for treatment of elevated blood ketones
- Participants will be required to have a home glucagon emergency kit. Participants who currently do not have one will be given a prescription for the glucagon emergency kit.

### 3.5 Assessment of Successful Completion of the Run-in Phase

- Enrolled participants will return approximately 14 days after the initiation of the run-in phase to assess progress or successful completion of the phase. If needed, one or more interim visits or
- phone contacts may occur to assist the participant with any system use issues. Visit procedures
- will include the following:

- Assessment of compliance with the use of either or both CGM and/or study pump (if applicable)
- Assessment of compliance with the use of:
- 670 CGM,
- o study pump,
- Assessment of skin reaction in areas where a CGM sensor was worn
- Assessment of eligibility to continue to the randomized control trial (RCT) phase of the study
- The appropriate study equipment will be downloaded and reviewed after the first 2 weeks of the
- run-in phase have been completed; participants will be evaluated for compliance and progress. If
- 677 that run-in phase occurred without any major safety issues, participants who are completing only
- the CGM run-in can be randomized. Those completing study pump and CGM may continue the
- run-in phase for another 2-4 weeks at PI discretion. In addition, MDI or study-pump naïve
- participants will be contacted by study staff within approximately 24hrs, 72hrs, and 1 week after
- pump initiation to answer any questions related to device use prior to the 2-week visit. All
- participants may have unlimited contact with the study team as needed.

- To enter the randomized trial from the run-in phase, participants must have obtained CGM
- readings on at least 11 out of the previous 14 days of the run-in phase (if applicable) and pump-
- naïve patients must have successfully used the study pump each day (if applicable). If a participant
- fails to meet either or both of these criteria, or if it is determined that the participant will benefit
- from additional time with equipment training, then the run-in period may be extended at the
- discretion of the investigator. One or two additional periods may occur, each a minimum of 11
- days with a goal of at least 14 days, with another clinic visit to assess results after each period
- using the same criteria as above. The run-in duration will therefore vary from approximately 2 to 6
- weeks, depending on the participant. Additional visits and phone contacts for further training are
- at investigator discretion.
- An assessment of CGM and pump knowledge will be made and the participant must demonstrate
- sufficient competency to proceed to the RCT. The trainer and participant will review the individual
- items listed on the pump training checklist to ensure competency.
- Participants who are unable to meet the CGM or study pump compliance requirements and those
- who no longer meet all of the inclusion and exclusion criteria will be withdrawn from the study.
- 698 If the participant is eligible to continue in the study, study staff will follow the procedure for insulin
- pump optimization described below in section 3.6.

## 3.6 Optimization of Insulin Pump Settings

- Data-driven optimization of pump settings will occur at the following times:
- For the first phase: Prior to Randomization:
- 703 O At the Run-in Review Visit
- Following Randomization visit and initiation of Extension Phase:
- 705 o If needed at the criteria of the physician at each clinical center, optimization may be done by phone contacts or in clinic visits.
- 707 o If the study participant contacts the study physician due to concerns about their pump settings due to recurring hypo- or hyperglycemia.
- 709 Data will be obtained from CGM and/or pump downloads at the visit. Adjustments to pump
- settings (basal rates, correction factor, insulin-to-carbohydrate ratio, etc.) will be made in response
- to major trends observed in the CGM data, with flexibility for clinicians to adhere to guidelines
- and practices established at each individual practice rather than a fixed set of heuristics for all
- 713 clinical centers.

## **Chapter 4: Randomization Visit**

#### 715 4.1 Randomization Visit

- The visit may occur on the same day as the Screening or Run-in Review Visit, or on a subsequent
- day. If deferred, the randomization visit should occur no more than 14 days after screening (if Run-
- 718 in skipped) or successful completion of the run-in phase.
- A urine pregnancy test will be repeated for all females of child-bearing potential if this visit is not
- on the same day as the Screening Visit.
- 721 **4.1.1 HbA1c**

- HbA1c will be measured using DCA Vantage or similar point-of-care (POC) device or local lab if
- this visit is not on the same day as the Screening Visit. A blood sample also will be drawn to send
- to the central laboratory for baseline HbA1c determination to be used in outcome analyses.
- 725 **4.1.2** Baseline C-Peptide Assessment
- A blood sample will be drawn to send to the central laboratory for a random, non-fasting C-peptide
- determination to characterize baseline residual insulin production. In conjunction, blood glucose
- may be measured using a blood glucose meter or a blood sample may be drawn to send to the
- 729 central laboratory for a blood glucose assessment.
- 730 **4.1.3 Randomization**
- 731 Eligible participants will be randomly assigned to one of two treatment groups in a 3:1 ratio:
- 732 1. Control-IQ Closed-Loop Control (CLC) Group
- 733 2. Standard of Care (SC) Group
- 734 The participant's randomization group assignment is determined by completing a Randomization
- Visit case report form on the study website. The randomization list will use a permuted block
- 736 design, stratified by clinical center.
- 737 The participant will be included in the data analysis regardless of whether or not the protocol for
- 738 the assigned randomization group is followed. Thus, the investigator must not randomize a
- 739 participant until he/she is convinced that the participant/parent will accept assignment to either
- 740 of the two groups.
- 741 It was decided that it was more important to stratify randomization by clinical center than by
- factors such as baseline time in range, HbA1c, or device use since these factors will be easier to
- adjust for in analysis than will clinical center in view of the relatively small number at each clinical
- 744 center.

## 745 **4.1.4 Questionnaires**

Participants will complete a set of baseline questionnaires, described in section 8.2 adapted for

747 age, prior to randomization.

## **Chapter 5: Main Study Procedures**

## 749 **5.1 Procedures for the CLC Group**

- 750 Participants assigned to the CLC group will receive study system training. These training
- sessions can occur on the same day or extend to up to one additional day if needed within 1-7
- days from randomization; participants will not take the study system home until training has
- been completed.

748

- 754 The parent/guardian will be trained on severe hypoglycemia emergency procedures including
- removal of the study pump and administration of glucagon. The parent/guardian will be asked to
- attend any/all of the other training procedures.

## 757 **5.2 Study System Training**

- 758 Participants will receive study system training by a qualified trainer. The study system includes
- 759 the Tandem t:slim X2 with Control-IQ technology and associated Dexcom G6 CGM.
- 760 CGM training will include:
- The participant will be instructed and supervised on how to insert the sensor and transmitter.
- The participant will learn how to calibrate the CGM unit
- The participant will learn how to access the CGM trace via the t:slim X2 with Control-IQ user interface
- Participants will be asked to perform fingerstick blood glucose measurements in accordance with the labeling of the study CGM device
- 767 Pump training will include:
- The participant will be fully instructed on the study insulin pump. A qualified system trainer will conduct the training and in particular discuss differences from their home pump in important aspects such as calculation of insulin on board and correction boluses. Additional topics not limited to but may include: infusion site initiation, cartridge/priming procedures, setting up the pump, charging the pump, navigation through menus, bolus procedures including stopping a bolus, etc.
- The study team will assist the participant in study pump infusion site initiation and will start the participant on the study pump. The study pump will be programmed with the participant's usual basal rates and pump parameters. The participant's personal pump will be removed.
- The participant will be supervised with the study pump during at least one meal or snack bolus to ensure participant understanding of the pump features.
- The participant will be encouraged to review the literature provided with the pump and infusion sets after the training is completed.
- Pump training specific to the Control-IQ Technology functions will include:
- How to turn on and off Control-IQ technology.
- How to understand when Control-IQ is increasing or decreasing basal rates.
- How to administer a meal or correction bolus on the t:slim X2 with Control-IQ system
- What to do when exercising while using the system
- How to enable the sleep function and set the sleep schedule
- The participant will be assessed for understanding of the system interface and how to react to safety/alert messages.
- The participant will be given a User Guide as a reference.

# 790 **5.2.1 System Initiation**

- 791 The participant will be instructed to use the system in closed-loop mode except 1) when no
- 792 calibrated CGM sensor is available or 2) if insulin is delivered by any means other than the
- study pump (e.g. injection of subcutaneous insulin via syringe in the event of infusion site failure).
- 794 If insulin is delivered by any means other than the study pump, participant will be instructed to
- 795 turn off Control-IQ for approximately four hours.
- The participant will also be instructed to contact study staff during periods of illness with an
- 797 elevated temperature >101.5 degrees Fahrenheit (38.6 degrees Celsius), periods of significant
- 798 illness, or during periods of use of medications such as epinephrine for the emergency treatment
- of a severe allergic reaction or asthma attack in addition to use of oral or injectable glucocorticoids
- to determine if closed-loop use should be temporarily discontinued.
- The participant's parent/legal guardian will be required to attend the training procedures and will
- be trained in all aspects aforementioned. All training will be conducted considering age of
- participant and parent involvement on diabetes treatment.
- Participants will be provided with sufficient supplies to last until the subsequent visit.
- Participants will be provided with contact information and will be asked to call the study
- 806 clinical staff for any health-related issues and for technical issues with t:slim X2 with
- 807 Control-IQ. Participants may use the study pump without Control-IQ activated and study
- 808 CGM during periods of component disconnections or technical difficulties. Participants will
- also receive study staff contact information to ask any questions they may have during the study.
- 810 Study staff will discuss with the participant that routine contact is required and will make
- arrangements with the participant for the contacts. If the participant cannot be reached, the
- participant's other contact methods will be utilized, including the emergency contact. Participants
- who are not compliant with the arranged contacts on two separate occasions may be discontinued
- at the discretion of the investigator.
- Upon completion of the t:slim X2 with Control-IQ training, study staff will document, using a
- checklist, that the participant is familiar with the function/feature and/or capable of performing
- each of the tasks specified.

- Participants will be provided Hypoglycemia, Hyperglycemia and Ketone Guidelines (section 7.2)
- for when their glucose levels are >300 mg/dL for more than two hours or >400 mg/dL at any time
- 820 or <70 mg/dL or ketones  $\ge$ 1.5 mmol/L.

# 5.2.2 Home Use of the Study System

- After training on the study system has been completed, participants will proceed with home use
- 823 (meaning free-living use at school, home, etc.) of the t:slim X2 with Control-IQ technology
- 824 system.
- Participants may use available manufacturer-provided software and features of the study CGM
- related to mobile data access or remote monitoring, but will be instructed not to use any third-party
- components for this purpose.

# 828 **5.2.3 Study Device Download**

- 829 Participants will be instructed to download the study device prior to each phone visit or on at least
- every 3-week basis throughout the remainder of the study.

#### **5.2.4 1-Week Phone Contact**

- Study staff will perform a phone call with the participant within 7 ( $\pm 1$ ) days following
- 833 randomization.
- 834 The following will occur:
- Assessment of compliance with study device use by review of any available device data
- Assessment of adverse events, adverse device effects, and device issues
- Study staff will answer any questions related to device use
- 838 Participants will then complete an additional week of home use with the study system. Participants
- will return to clinic 14 ( $\pm$ 3) days from the date of randomization.

### 5.2.5 2-Week Visit (Training Review and Insulin Pump Optimization)

- The participant will be offered review training to address any questions on the use of the study
- device including meal bolus strategies and strategies related to pump use and exercise.
- 843 The following will occur:
- Assessment of compliance with study device use by review of any available device data
- Assessment of adverse events, adverse device effects, and device issues
- Study staff will answer any questions related to device use and follow the procedure for insulin
- pump optimization described in section 3.6 using the study CGM available data from the
- previous two weeks.
- The blood glucose meter and study ketone meter will be downloaded and QC tested with control solution.

## **5.3 Procedures for the SC Group**

- Participants in the SC group will use an insulin pump that they usually use for the treatment of
- their diabetes or a study pump provided by the study team if they are transitioning from MDI to
- pump for the study, in conjunction with the study CGM, study blood glucose meter, and study
- ketone meter. Study pump training and/or study CGM training will be provided if the participant
- is initiating use of these devices at this point.
- 857 If a participant is using a pump with a LGS feature, he/she will be allowed to continue using this
- 858 feature during the trial.
- Participants may use available manufacturer-provided software and features of the study CGM
- related to mobile data access or remote monitoring, but will be instructed not to use any third-party
- components for this purpose.

# 862 5.3.1 Study Device Data Download

- Participants will be instructed to upload data from the study CGM using commercially available
- software prior to the 1-week phone contact and prior to the 2-week clinic visit for clinician review.
- Participants will be provided with any software and hardware needed to perform these data
- wploads.

#### 867 5.3.2 1-Week Phone Contact

- Study staff will perform a phone call with the participant  $7(\pm 1)$  days following randomization.
- 869 The following will occur:
- Assessment of compliance with study device use by review of any available device data
- Assessment of adverse events, adverse device effects, and device issues
- Study staff will answer any questions related to device use
- The participant will continue on SC for a second week, then return to the clinic 14 ( $\pm$ 3) days from
- 874 the date of randomization.

# 875 5.3.3 2-Week Visit (Training Review and Insulin Pump Optimization)

- The participant will be offered review training on the use of SC during the remainder of the study,
- including meal bolus strategies and strategies related to pump use and exercise.
- 878 The following will occur:
- Assessment of compliance with study device use by review of any available device data
- Assessment of adverse events, adverse device effects, and device issues
- Study staff will review uploaded CGM data, answer any questions related to device use, and follow the procedure for insulin pump optimization described in section 3.6.
- The study blood glucose meter and study ketone meter will be downloaded and QC tested with

- 884 at least two different concentrations of control solution if available.
- 885 The participant will be instructed to upload data from the CGM at least once every 4 weeks for the
- 886 remainder of the study.

#### 887 5.4 Follow-up Visits and Phone Contacts for Both Groups

- 888 The schedule for remaining follow-up visits and phone contacts is the same for both treatment
- groups. Study staff will discuss with the participant that periodic contact is required and will make 889
- 890 arrangements with the participant for the contacts. If the participant or parent/guardian, cannot be
- 891 reached, the participant's other contact methods will be utilized, including the emergency contact.

#### 892 5.4.1 Follow-up Visits

- 893 Follow-up visits in clinic will occur at:
- 894 2 week ( $\pm 3$  days)

897

- 895 • 8 weeks ( $\pm 1$  week)
- 896 • 16 weeks (+1 week) – end of Main Study Phase

#### **5.4.1.1 Procedures at Follow-up Visits**

- 898 Procedures performed in both groups at each visit, unless otherwise specified below:
- 899 Assessment of compliance with study device use by review of any available device data
- 900 Assessment of adverse events, adverse device effects, and device issues
- 901 Download of device data (study system or personal pump and study CGM, study BG meter, 902 study ketone meter)

#### 903 **5.4.2 Phone Contacts**

- In addition to the 1-week phone contact described above for the respective treatment groups, the 904
- 905 following phone contacts will be made:
- 906 • 4 weeks ( $\pm 3$  days)
- 907 • 6 weeks ( $\pm 3$  days)
- 908 • 10 weeks (±3 days)
- 909 • 12 weeks (±3 days)
- 910 • 14 weeks (±3 days)
- 911 At each phone contact, the following procedures are performed in both treatment groups:
- 912 Review of available CGM and/or system data to identify any safety issues associated with 913 insulin pump settings and current diabetes management approach
- 914 Assessment of adverse events, adverse device effects, and device issues

- Additional phone contacts may be performed as needed.
- 916 **5.4.3 Data from Study Devices**
- All participants will be asked to upload data from the CGM at least once every 4 weeks during the
- 918 extension phase. The study staff will confirm that the data were received.
- 919 5.4.4 16-Week Final First Phase Visit
- All participants will return to the clinic for a 16-Week (+7 days) final clinic visit during which the
- 921 following will occur:
- HbA1c determination using the DCA Vantage or similar point of care device
- Collection of a blood sample to send to the central laboratory for HbA1c determination
- Completion of questionnaires
- Weight and height measurement will be repeated
- Assessment of adverse events, adverse device effects, and device issues
- Download of device data (study system or personal pump and study CGM, study BG meter, study ketone meter)
- 929 **5.5 Early Termination Visit (If Applicable)**
- Participants will be asked to come for an end of study visit in the event of withdrawal or early
- 931 termination.
- 932 **5.6** Unscheduled Visits
- 933 Participants may have unscheduled visits during the study period if required for additional device
- training or other unanticipated needs per the study investigator discretion.
- 935 5.7 Participant Access to Study Device at Study Closure
- Participant will return all investigational study devices and supplies (insulin pump, CGM and
- 937 related supplies) at study closure. Participant may keep the study ketone meter and study
- glucometer if these devices are not marked for investigational use only.

# **Chapter 6: Extension Phase Procedures**

- At the conclusion of the 16-week visit, all participants will have the option to use of the Control-
- 941 IQ closed-loop system.

939

- 942 6.1 Closed Loop Control Participants
- Participants who have completed the 16-week Main Study Phase will be provided the option to
- ontinue the use the t:slim with Control-IQ System for an additional 12 weeks.
- The following phone contacts will be made for CLC Group participants in the Extension Phase:
- 946 20 week (±3 days)
- 947 24 week (±3 days)
- 948 At each phone contact, the following procedures are performed:
- Review of available CGM and/or system data to identify any safety issues associated with insulin
- pump settings and current diabetes management approach
- Assessment of adverse events, adverse device effects, and device issues
- 952 **6.2 SC Group Participants**
- 953 Training on pump (section 5.2) use will be provided and therapy optimization will occur as
- 954 follows:
- If needed at the criteria of the physician at each clinical center, optimization may be done at either phone contacts or in clinic visits.
- If the study participant contacts the study physician due to concerns about their pump settings due to recurring hypo- or hyperglycemia.
- 959 Data will be obtained from CGM and/or pump downloads at the visit. Adjustments to pump
- settings (basal rates, correction factor, insulin-to-carbohydrate ratio, etc.) will be made in response
- to major trends observed in the CGM data, with flexibility for clinicians to adhere to guidelines
- and practices established at each individual practice rather than a fixed set of characteristics for all
- 963 clinical centers.
- The following phone contacts will be made for SC Group participants in the Extension Phase:
- 965 17 weeks (±3 days)
- 966 19 weeks (±3 days)
- 967 21 weeks (±3 days)

- 968 25 weeks (±3 days)
- At each phone contact, the following procedures are performed:
- Review of available CGM and/or system data to identify any safety issues associated with insulin pump settings and current diabetes management approach
- Assessment of adverse events, adverse device effects, and device issues
- 973 Follow-up visits for SC group during the Extension Phase in clinic will occur at:
- 974 23 Weeks (±1 week)
- 975 28 Weeks (+1 week) End of Study
- 976 Procedures Specific to the 28 Week Visit
- HbA1c determination using the DCA Vantage or similar point of care device
- Collection of a blood sample to send to the central laboratory for HbA1c determination
- Completion of questionnaires
- Weight measurement will be repeated, in addition to height
- Insulin Pump Optimization as described above
- 982 **6.3** Early Termination Visit (If Applicable)
- 983 Participants will be asked to come for an end of study visit in the event of withdrawal or early
- 984 termination.
- 985 **6.4 Unscheduled Visits**
- 986 Participants may have unscheduled visits during the study period if required for additional device
- training or other unanticipated needs per the study investigator discretion.
- 988 6.5 Participant Access to Study Device at Study Closure
- 989 Participant will return all investigational study devices and supplies (insulin pump, CGM and
- 990 related supplies) at study closure. Participant may keep the study ketone meter and study
- glucometer if these devices are not marked for investigational use only.

# 992 Chapter 7: Study Devices

- 993 7.1 Description of the Investigational Device
- 994 **7.1.1 Insulin Pump**
- The study system will include the Tandem t:slim X2 with Control-IQ technology.
- 996 7.1.2 Continuous Glucose Monitoring
- 997 The study CGM will include Dexcom G6 transmitter and sensors when using the Tandem t:slim
- 998 X2 with Control-IQ technology. This may not be an FDA-approved device system at the start of
- 999 the study, but may become approved during the course of the study. The CGM sensor will be
- replaced at least once every 10 days.
- 1001 7.1.3 Blood Glucose Meter and Strips
- Blood glucose levels will be measured using the study's blood glucose meter (glucometer) and the
- 1003 CGM device will be calibrated if needed using the study glucometer and strips in accordance with
- the manufacturer's labeling.
- 1005 7.1.4 Ketone Meter and Strips
- 1006 Blood ketone levels will be measured using the Abbott Precision Xtra meter and strips in
- accordance with the manufacturer's labeling. The blood glucose meter component of the Precision
- 1008 Xtra device will not be used.
- 1009 7.1.5 Study Device Accountability Procedures
- Device accountability procedures will be detailed in the clinical center procedures manual.
- 1011 **7.1.6 Blood Ketone Testing**
- Participants to perform QC testing at home per manufacturer guidelines.
- All study blood ketone meters will be QC tested with control solution if available during all
- office visits. A tested meter will not be used in a study if it does not read within the target
- range at each concentration per manufacturer labeling. The participant will be instructed to
- contact study staff for a replacement of the meter, test strips, and control solution if a meter
- fails QC testing at home.
- Participants will be instructed on how to perform blood ketone testing.
- Participants will be given guidelines for treatment of elevated blood ketones.
- 1020 **7.2 Safety Measures**
- **7.2.1 CGM Calibration**
- Throughout the study, participants will be instructed to calibrate the study CGM in accordance
- with manufacturer labelling.

# **7.2.2 System Failure**

- 1025 If the CGM signal becomes unavailable for more than 20 minutes consecutively, Control-IQ or
- 1026 closed loop will not operate to automatically adjust insulin. If the CGM is not connected, the
- system will revert to usual function of the pump and deliver insulin with the insulin dosing
- parameters programmed in the system for that individual. Resumption of Closed-Loop will
- occur automatically once CGM signal is available again.
- 1030 If the study system is unable to activate Control-IQ for any reason, the pump will automatically
- revert to preprogrammed basal insulin delivery without any need for instruction from the user.
- 1032 If the t:slim X2 detects a system error that does not allow the pump to operate, the Malfunction
- Alarm will display and the participant will be instructed to contact Tandem Technical Support via
- the study team.

# 1035 7.2.3 Hypoglycemia Threshold Alert and Safety Protocol

- During the course of the study, participants will be permitted to change the CGM low glucose
- threshold alert setting on their device or mobile app, but will be instructed to choose a value no
- less than 70 mg/dL.
- The t:slim X2 with Control-IQ system will issue a predictive hypoglycemia alert (Control-IQ Low
- 1040 Alert) when the system predicts BG <70 mg/dL within the next 15 minutes (<80 mg/dL when
- 1041 exercise mode is activated).
- 1042 If the participant receives a Control-IQ Low Alert, a message appears on the user interface (UI)
- that is accompanied by vibration followed by vibrations and/or sound if not acknowledged by the
- user in 5 minutes. This alert remains on the screen until acknowledged by the user. The user is
- prompted to test blood sugar and treat with carbs.

#### 1046 7.2.4 Hyperglycemia Threshold Alert and Safety Protocol

- During the course of the study, participants will be permitted to change the CGM high glucose
- threshold alert setting on their device or mobile app, but will be instructed to choose a value no
- 1049 greater than 300 mg/dL.
- The t:slim X2 with Control-IQ system will issue a predictive hyperglycemia alert (Control-IQ
- High Alert) when the system has increased insulin delivery, but detects a CGM value above 200
- 1052 mg/dL and does not predict the value will decrease in the next 30 minutes.
- 1053 If the participant receives a Control-IQ High Alert, a message appears on the UI that is
- accompanied by vibration followed by vibrations and/or sound if not acknowledged by the user in
- 5 minutes. This alert remains on the screen until acknowledged by the user. The user is prompted
- to check the site for occlusion and test blood glucose.
- 1057 If a participant's CGM reading is >300 mg/dL for over 2 hours or ≥400 mg/dL at any point, the
- participant will be instructed to take the following steps:
- Perform a blood glucose meter check.

- If the blood glucose is >300 mg/dL, check for blood ketones with the study ketone meter.
- If the ketone level is ≥1.5 mmol/L, take correction insulin, change insulin (pump) infusion site and contact study staff.
- If a participant administers correction insulin via insulin syringe, participants will be instructed to turn Control-IQ off for approximately four hours.

# **Chapter 8: Testing Procedures and Questionnaires**

- 1066 **8.1 Laboratory Testing**
- 1067 **8.1.1 Comprehensive Metabolic Panel (CMP)**
- 1068 A blood sample will be obtained at screening to assess kidney and liver functioning.
- 1069 **8.1.2 HbA1c**:

1065

- Performed locally at the Screening visit, Randomization visit and the 16-week visit.
- A blood sample will be obtained and sent to central lab at the Randomization visit, at the 16week visit and at the end of the study visit.
- **8.1.3 Urine Pregnancy:**
- 1074 Performed locally for females of child-bearing potential at the Screening visit and the
- Randomization visit. This will also be done anytime pregnancy is suspected.
- 1076 **8.1.4 C-peptide and Glucose**
- 1077 Blood samples will be obtained and sent to the central lab at the Randomization visit. Back-up
- samples will be stored on-site until all samples are resulted.
- 1079 **8.2 Questionnaires**
- 1080 Questionnaires are completed at the Randomization Visit and Week 16 Visit for all participants.
- Participants who complete the Extension Phase will also complete the questionnaires at Week 28.
- The questionnaires will be family and age appropriate are described briefly below. The procedures
- for administration are described in the clinical center procedures manual.
- The following questionnaires will be completed at the Randomization Visit:
- Clarke's Hypoglycemia Awareness Scale Child and Parent (Children age 10+ years at the time of consent will complete as well as all Parents)
- Fear of Hypoglycemia Survey (HFS-II) Child and Parent
- Problem Areas In Diabetes Survey (PAID) Child and Parent
- Pediatric Quality of Life Child and Parent
- INSPIRE Survey Child and Parent
- Pittsburgh Sleep Quality Index (PSQI) Parent
- The following questionnaires will be completed at the Week 16 and Week 28 Visits:
- Clarke's Hypoglycemia Awareness Scale Child and Parent (Children age 10+ years at the time of consent will complete as well as all Parents)

- Fear of Hypoglycemia Survey (HFS-II) Child and Parent
- Problem Areas In Diabetes Survey (PAID) Child and Parent
- Pediatric Quality of Life Child and Parent
- INSPIRE Post-Assessment Survey Child and Parent
- Pittsburgh Sleep Quality Index (PSQI) Parent
- System Usability Scale (SUS) Closed-Loop participants only
- Administration time is approximately 15 minutes.

# 8.2.1 Clarke's Hypoglycemia Awareness Scale – Child and Parent

- The scale comprises eight questions characterizing the participant's exposure to episodes
- of moderate and severe hypoglycemia. It also examines the glycemic threshold for, and
- symptomatic responses to hypoglycemia. A score of four or more on a scale of 0 to 7 implies
- impaired awareness of hypoglycemia.
- Administration time is approximately 5 minutes.

# 1108 8.2.2 Hypoglycemia Fear Survey (HFS-II)/Low Blood Sugar Survey – Child and Parent

- The Hypoglycemia Fear Survey-II was developed to measure behaviors and worries related to fear
- of hypoglycemia in adults with type 1 diabetes. It is composed of 2 subscales, the Behavior (HFS-
- B) and Worry (HFS-W). HFS-B items describe behaviors in which patients may engage to avoid
- hypoglycemic episodes and/or their negative consequences (e.g., keeping blood glucose levels
- higher, making sure other people are around, and limiting exercise or physical activity). HFS-W
- items describe specific concerns that patients may have about their hypoglycemic episodes (e.g.,
- being alone, episodes occurring during sleep, or having an accident). HFS-II was adapted for
- children and parents. Items are rated on a 5-point Likert scale (0=never, 4=always), with higher
- scores indicating higher fear of hypoglycemia.
- Administration time is approximately 10 minutes (both versions).

### 8.2.3 Problem Areas In Diabetes Survey (PAID) – Child and Parent

- The Problem Areas In Diabetes Survey is a measure of diabetes-related emotional distress and
- 1121 consists of a scale of 16 items for the Parent version and 11 items for the Child version. Patients
- and parents rate the degree to which each item is currently problematic for them on a 6-point Likert
- scale, from 1 (no problem) to 6 (serious problem).
- 1124 Administration time is approximately 10 minutes.

#### 1125 **8.2.4 PedsQL Diabetes Module – Child and Parent**

- This is a 33-item scale developed and validated for the measurement of diabetes-specific quality
- of life. Separate forms have been validated for child self-report (5-7 year old; 8-12 year old; and
- 1128 12-18 year old) and parent report for these same age groups. Participants record the extent to

- which they (or their child) experienced each of 33 problems related to diabetes in the prior
- 1130 month.
- Administration time is approximately 15 minutes.
- 1132 8.2.5 INSPIRE Survey Child and Parent
- 1133 The INSPIRE (Insulin Delivery Systems: Perceptions, Ideas, Reflections and Expectations) survey
- was developed to assess various aspects of a user's experience regarding automated insulin
- delivery for both patients and family members. The surveys include various topics important to
- patients with type 1 diabetes and their family members based upon >200 hours of qualitative
- interviews and focus groups. The child pre-assessment survey includes 27 items, and the parent
- pre-assessment survey includes 45 items. The post-assessment child survey includes 17 items, and
- the parent post-assessment contains 21 items. Response options for all surveys include a 5-point
- Likert scale from strongly agree to strongly disagree, along with an N/A option.
- 1141 Administration time is approximately 5 minutes.
- 8.2.6 Pittsburgh Sleep Quality Index (PSQI) Parent
- Pittsburgh Sleep Quality Index (PSQI) is a 10-item questionnaire that measures the sleep quality
- and pattern of sleep in adults. Seven component scores are derived, each scored 0 (no difficulty)
- to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to
- 1146 21). Higher scores indicate worse sleep quality.
- 1147 Administration time is approximately 5 minutes.
- 1148 8.2.7 System Usability Scale (SUS) Closed-Loop participants only
- The System Usability Scale (SUS) is a 10-item questionnaire that measures the overall usability of
- a system. It is a valid and reliable measure of the perceived usability of a system and is technology-
- agnostic. The questionnaire presents statements with five response options (anchoring the options
- from strongly disagree to strongly agree) and asks users to rate their agreement to the statements.
- User scores are transformed into a composite score, from 0 to 100, and this score is taken as an
- overall measure of the system's usability; higher scores indicate better perceived usability.
- 1155 Administration time is approximately 5 minutes.

# 1156 Chapter 9: Adverse Events, Device Issues, and Stopping Rules

- 1157 **9.1 Adverse Events**
- 1158 **9.1.1 Definitions**
- Adverse Event (AE): Any untoward medical occurrence in a study participant, irrespective of the
- relationship between the adverse event and the device(s) under investigation (see section 9.1.2 for
- reportable adverse events for this protocol).
- 1162 <u>Serious Adverse Event (SAE):</u> Any untoward medical occurrence that:
- 1163 Results in death.
- Is life-threatening; (a non-life-threatening event which, had it been more severe, might have become life-threatening, is not necessarily considered a serious adverse event).
- Requires inpatient hospitalization or prolongation of existing hospitalization.
- Results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions (sight threatening).
- Is a congenital anomaly or birth defect.
- Is considered a significant medical event by the investigator based on medical judgment (e.g., may jeopardize the participant or may require medical/surgical intervention to prevent one of the outcomes listed above).
- 1173 <u>Unanticipated Adverse Device Effect (UADE):</u> Any serious adverse effect on health or safety or
- any life-threatening problem or death caused by, or associated with, a device, if that effect,
- problem, or death was not previously identified in nature, severity, or degree of incidence in the
- investigational plan or application (including a supplementary plan or application), or any other
- unanticipated serious problem associated with a device that relates to the rights, safety, or welfare
- 1178 of participants (21 CFR 812.3(s)).
- 1179 Adverse Device Effect (ADE): Any untoward medical occurrence in a study participant which the
- device may have caused or to which the device may have contributed (Note that an Adverse Event
- Form is to be completed in addition to a Device Deficiency or Issue Form).
- Device Complaints and Malfunctions: A device complication or complaint is something that
- happens to a device or related to device performance, whereas an adverse event happens to a
- participant. A device complaint may occur independently from an AE, or along with an AE.
- An AE may occur without a device complaint or there may be an AE related to a device complaint.
- 1186 A device malfunction is any failure of a device to meet its performance specifications or otherwise
- perform as intended. Performance specifications include all claims made in the labeling for the
- device. The intended performance of a device refers to the intended use for which the device is
- labeled or marketed. (21 CFR 803.3). Note: for reporting purposes, clinical centers will not be
- asked to distinguish between device complaints and malfunctions.

# 1191 **9.1.2 Reportable Adverse Events**

- For this protocol, a reportable adverse event includes any untoward medical occurrence that meets
- one of the following criteria:
- 1. A serious adverse event

1205

1216

- 2. An Adverse Device Effect as defined in section 9.1.1, unless excluded from reporting in section 9.2
- 3. An Adverse Event occurring in association with a study procedure
- 1198 4. Hypoglycemia meeting the definition of severe hypoglycemia as defined below
- 5. Diabetic ketoacidosis (DKA) as defined below or in the absence of DKA, a hyperglycemic or ketosis event meeting the criteria defined below
- Hypoglycemia and hyperglycemia not meeting the criteria below will not be recorded as adverse
- events unless associated with an Adverse Device Effect. Skin reactions from sensor placement are
- only reportable if severe and/or required treatment.
- Pregnancy occurring during the study will be recorded.

## 9.1.2.1 Hypoglycemic Events

1206 Hypoglycemia not associated with an Adverse Device Effect is only reportable as an adverse event 1207 when the following definition for severe hypoglycemia is met: the event required assistance of another person due to altered consciousness, and required another person to actively administer 1208 1209 carbohydrate, glucagon, or other resuscitative actions. This means that the participant was impaired cognitively to the point that he/she was unable to treat himself/herself, was unable to 1210 1211 verbalize his/ her needs, was incoherent, disoriented, and/or combative, or experienced seizure or 1212 coma. These episodes may be associated with sufficient neuroglycopenia to induce seizure or 1213 coma. If plasma glucose measurements are not available during such an event, neurological 1214 recovery attributable to the restoration of plasma glucose to normal is considered sufficient 1215 evidence that the event was induced by a low plasma glucose concentration.

#### 9.1.2.2 Hyperglycemic Events/Diabetic Ketoacidosis

- Hyperglycemia not associated with an Adverse Device Effect is only reportable as an adverse event when one of the following 4 criteria is met:
- the event involved DKA, as defined by the Diabetes Control and Complications Trial (DCCT) and described below
- evaluation or treatment was obtained at a health care provider facility for an acute event involving hyperglycemia or ketosis
- blood ketone level ≥1.5 mmol/L and communication occurred with a health care provider at
   the time of the event
- blood ketone level ≥3.0 mmol/L, even if there was no communication with a health care provider

- Hyperglycemic events are classified as DKA if the following are present:
- Symptoms such as polyuria, polydipsia, nausea, or vomiting;
- Serum ketones ≥1.5 mmol/L or large/moderate urine ketones;
- Either arterial blood pH <7.30 or venous pH <7.24 or serum bicarbonate <15; and
- Treatment provided in a health care facility
- 1232 All reportable Adverse Events—whether volunteered by the participant, discovered by study
- personnel during questioning, or detected through physical examination, laboratory test, or other
- means—will be reported on an adverse event form online. Each adverse event form is reviewed
- by the Medical Monitor to verify the coding and the reporting that is required.

# 1236 9.1.3 Relationship of Adverse Event to Study Device

- The study investigator will assess the relationship of any adverse event to be related or unrelated
- by determining if there is a reasonable possibility that the adverse event may have been caused by
- the study device.
- 1240 To ensure consistency of adverse event causality assessments, investigators should apply the
- following general guideline when determining whether an adverse event is related:
- 1242 <u>Yes</u>
- There is a plausible temporal relationship between the onset of the adverse event and the study
- intervention, and the adverse event cannot be readily explained by the participant's clinical state,
- intercurrent illness, or concomitant therapies; and/or the adverse event follows a known pattern of
- response to the study intervention; and/or the adverse event abates or resolves upon discontinuation
- of the study intervention or dose reduction and, if applicable, reappears upon re-challenge.
- 1248 No
- Evidence exists that the adverse event has an etiology other than the study intervention (e.g.,
- 1250 preexisting medical condition, underlying disease, intercurrent illness, or concomitant
- medication); and/or the adverse event has no plausible temporal relationship to study intervention.

### 1252 9.1.4 Intensity of Adverse Event

- The intensity of an adverse event will be rated on a three point scale: (1) mild, (2) moderate, or (3)
- severe. It is emphasized that the term severe is a measure of intensity: thus, a severe adverse event
- is not necessarily serious. For example, itching for several days may be rated as severe, but may
- not be clinically serious.
- MILD: Usually transient, requires no special treatment, and does not interfere with the participant's daily activities.
- MODERATE: Usually causes a low level of inconvenience or concern to the participant and may interfere with daily activities, but is usually ameliorated by simple therapeutic measures.

• SEVERE: Interrupts a participant's usual daily activities and generally requires systemic drug therapy or other treatment.

# 1263 9.1.5 Coding of Adverse Events

- 1264 Adverse events will be coded using the MedDRA dictionary. The Medical Monitor will review
- the investigator's assessment of causality and may agree or disagree. Both the investigator's and
- Medical Monitor's assessments will be recorded. The Medical Monitor will have the final say in
- determining the causality.
- Adverse events that continue after the participant's discontinuation or completion of the study will
- be followed until their medical outcome is determined or until no further change in the condition
- is expected.

#### 1271 9.1.6 Outcome of Adverse Event

- 1272 The outcome of each reportable adverse event will be classified by the investigator as follows:
- RECOVERED/RESOLVED The participant recovered from the AE/SAE without sequelae.

  Record the AE/SAE stop date.
- RECOVERED/RESOLVED WITH SEQUELAE The event persisted and had stabilized without change in the event anticipated. Record the AE/SAE stop date.
- FATAL A fatal outcome is defined as the SAE that resulted in death. Only the event that was the cause of death should be reported as fatal. AEs/SAEs that were ongoing at the time of death; however, were not the cause of death, will be recorded as "resolved" at the time of death.
- NOT RECOVERED/NOT RESOLVED (ONGOING) An ongoing AE/SAE is defined as the event was ongoing with an undetermined outcome.
- 1282 O An ongoing outcome will require follow-up by the clinical center in order to determine the final outcome of the AE/SAE.
- 1284 o The outcome of an ongoing event at the time of death that was not the cause of death, will be updated and recorded as "resolved" with the date of death recorded as the stop date.
- UNKNOWN An unknown outcome is defined as an inability to access the participant or the participant's records to determine the outcome (for example, a participant that was lost to follow-up).
- 1289 All clinically significant abnormalities of clinical laboratory measurements or adverse events
- 1290 occurring during the study and continuing at study termination should be followed by the
- participant's physician and evaluated with additional tests (if necessary) until diagnosis of the
- underlying cause, or resolution. Follow-up information should be recorded on source documents.
- 1293 If any reported adverse events are present when a participant completes the study, or if a participant
- is withdrawn from the study due to an adverse event, the participant will be contacted for re-
- evaluation within 2 weeks. If the adverse event has not resolved, additional follow-up will be
- performed as appropriate. Every effort should be made by the Investigator or delegate to contact
- the participant until the adverse event has resolved or stabilized.

# 1298 **9.2 Reportable Device Issues**

- 1299 All UADEs, ADEs, device complaints, and device malfunctions will be reported irrespective of
- whether an adverse event occurred, except in the following circumstances.
- The following device issues are anticipated and will not be reported on a Device Issue Form but
- will reported as an Adverse Event if the criteria for AE reporting described above are met:
- Component disconnections
- CGM sensors lasting fewer than the number of days expected per CGM labeling
- CGM tape adherence issues
- Pump infusion set occlusion not leading to ketosis
- Battery lifespan deficiency due to inadequate charging or extensive wireless communication
- Intermittent device component disconnections/communication failures not leading to system replacement
- Device issues clearly addressed in the user guide manual that do not require additional troubleshooting
- Skin reactions from CGM sensor placement or pump infusion set placement that do not meet criteria for AE reporting

## 1314 9.3 Pregnancy Reporting

- 1315 If pregnancy occurs, the participant will be discontinued from the study. The occurrence of
- pregnancy will be reported on an AE Form.

# 1317 **9.4 Timing of Event Reporting**

- 1318 SAEs and UADEs must be reported to the Coordinating Center within 24 hours via completion of
- the online serious adverse event form.
- Other reportable adverse events, device malfunctions (with or without an adverse event), and
- device complaints should be reported promptly by completion of an electronic case report form,
- but there is no formal required reporting period.
- 1323 The Coordinating Center will notify all participating investigators of any adverse event that is
- serious, related, and unexpected. Notification will be made within 10 days after the Coordinating
- 1325 Center becomes aware of the event.
- Each principal investigator is responsible for reporting serious study-related adverse events and
- abiding by any other reporting requirements specific to his/her Institutional Review Board or
- 1328 Ethics Committee.
- Upon receipt of a UADE report, the Sponsor will investigate the UADE and if indicated, report
- the results of the investigation to the clinical centers' IRBs, and the FDA within 10 working days
- of the Sponsor becoming aware of the UADE per 21CFR 812.46(b). The Medical Monitor must
- determine if the UADE presents an unreasonable risk to participants. If so, the Medical Monitor
- must ensure that all investigations, or parts of investigations presenting that risk, are terminated as

- soon as possible but no later than 5 working days after the Medical Monitor makes this
- determination and no later than 15 working days after first receipt notice of the UADE.
- In the case of a device system component malfunction (e.g. pump, CGM, control algorithm),
- information will be forwarded to the responsible company by the clinical center personnel, to be
- handled by its complaint management system.

# 1339 9.5 Stopping Criteria

1340

### 9.5.1 Participant Discontinuation of Study Device

- Rules for discontinuing study device use are described below.
- The investigator believes it is unsafe for the participant to continue on the intervention. This
- 1343 could be due to the development of a new medical condition or worsening of an existing
- 1344 condition; or participant behavior contrary to the indications for use of the device that imposes
- on the participant's safety
- The participant requests that the treatment be stopped
- Participant pregnancy
- Two distinct episodes of DKA
- Two distinct severe hypoglycemia events as defined in section 9.1.2.1
- 1350 If pregnancy occurs, the participant will be discontinued from the study entirely. Otherwise, even
- if the study device system is discontinued, the participant will be encouraged to remain in the study
- through the final study visit.

#### 1353 9.5.2 Criteria for Suspending or Stopping Overall Study

- In the case of an unanticipated system malfunction resulting in a severe hypoglycemia or severe
- hyperglycemia event (as defined in section 9.1.2.2), use of the study device system will be
- suspended while the problem is diagnosed.
- In addition, study activities could be similarly suspended if the manufacturer of any constituent
- study device requires stoppage of device use for safety reasons (e.g. product recall). The affected
- study activities may resume if the underlying problem can be corrected by a protocol or system
- modification that will not invalidate the results obtained prior to suspension. The study Medical
- Monitor will review all adverse events and adverse device events that are reported during the study
- and will review compiled safety data at periodic intervals (generally timed to the review of
- compiled safety data by the DSMB). The Medical Monitor may request suspension of study
- activities or stoppage of the study if deemed necessary based on the totality of safety data available.

# 1365 9.6 Independent Safety Oversight

- 1366 A Data and Safety Monitoring Board (DSMB) will review compiled safety data at periodic
- intervals (typically every 6 months). In addition, the DSMB will review all DKA and severe
- hypoglycemia irrespective of relatedness to study device use, and all serious events (including
- UADEs) related to study device use at the time of occurrence. The DSMB also will be informed
- of any ADEs not meeting criteria for a UADE if the Medical Monitor requests the DSMB

- review. The DSMB can request modifications to the study protocol or suspension or outright
- stoppage of the study if deemed necessary based on the totality of safety data available. Details
- regarding DSMB review will be documented in a separate DSMB document.
- 1374 **9.7** Risks
- The potential risks associated with use of the study device are described in section 1.3.
- 1376 Additional risks are minor and/or infrequent and include:
- Pain, bruising, redness, or infection from blood draws
- 1378 Loss of confidentiality
- Stress from completing quality of life questionnaires

#### **Chapter 10: Miscellaneous Considerations** 1380 1381 10.1 Drugs Used as Part of the Protocol 1382 Participants will use either lispro or aspart insulin prescribed by their personal physician. 1383 10.2 Prohibited Medications, Treatments, and Procedures 1384 Participants using glulisine at the time of enrollment will be asked to contact their personal 1385 physician to change their prescribed personal insulin to lispro or aspart for the duration of the trial 1386 in the case they are randomized to experimental arm 1387 Treatment with any non-insulin glucose-lowering agent (including GLP-1 agonists, Symlin, DPP-1388 4 inhibitors, SGLT-2 inhibitors, biguanides, sulfonylureas and naturaceuticals) will not be 1389 permitted. 1390 The investigational study devices (t:slim X2 insulin pump, study CGM systems) must be removed 1391 before Magnetic Resonance Imaging (MRI), Computed Tomography (CT) or diathermy treatment. 1392 Participants may continue in the trial after temporarily discontinuing use if requiring one of the 1393 treatments above. 1394 10.3 Participant Withdrawal 1395 Participation in the study is voluntary, and a participant may withdraw at any time. For participants who withdraw, their data will be used up until the time of withdrawal. 1396 1397 **10.4 Confidentiality** 1398 For security and confidentiality purposes, participants will be assigned an identifier that will 1399 be used instead of their name. Protected health information gathered for this study will be 1400 shared with the coordinating center, the Jaeb Center for Health Research in Tampa, FL.

De-identified participant information may also be provided to research sites involved in the study.

De-identified participant information may also be provided to Tandem for system evaluation

1401

1402

1403

purposes.

# **Chapter 11: Statistical Consideration**

# 1405 11.1 Statistical and Analytical Plans

- 1406 The outcome metrics and the statistical analyses are summarized below. A detailed statistical
- analysis plan will be written and finalized prior to the first tabulation of data by treatment group
- 1408 (ie, for DSMB review). The analysis plan synopsis in this chapter contains the framework of the
- anticipated final analysis plan.

1404

## 1410 **11.2 Statistical Hypotheses**

- 1411 This study is an extension to children ages 6-13 years old, of the Main Protocol described in IDE
- 1412 G180053, which includes N=168 children ages 14 and up and adults. Thus, the primary outcome
- 1413 for this study is identical to the Main protocol CGM-measured % in range 70-180 mg/dL.
- 1414 The hypotheses for the primary outcome are:
- a. *Null Hypothesis*: There is no difference in mean CGM-measured % in range 70-180 mg/dL over 16 weeks between SC and CLC
- b. *Alternative Hypothesis*: The mean CGM-measured % in range 70-180 mg/dL over 16 weeks is different for SC and CLC.

# **14**19 **11.3 Sample Size**

- Sample size has been computed for the primary outcome (CGM-measured % in range 70-180
- mg/dL). Data from IDE G170267; Device Name: t:slim X2 with Control-IQ Technology; "Real-
- 1422 Time Monitoring and Glucose Control During Winter-Sport Exercise in Youth with Type 1
- Diabetes: The AP Ski Camp Continued" were used to calculate sample size specific to this age
- group. In this study, which was completed in the winter of 2018, 24 school-aged children (6-12)
- 1425 years) with type 1 diabetes participated in a 3-day ski camp (~5 h skiing/day), followed by an
- additional 72 hour at-home phase under parental supervision. Study participants were randomized
- 1427 1:1 to SAP and t:slim X2 with Control-IQ Technology. The data from the 72-hour home phase
- 1127 1.1 to 511 and 1.5111 1.12 with control of reemfology. The data from the 72 hour nome phase
- 1428 was used for this sample size calculation note that the closed-loop control system and the age
- range of the participants are identical to those proposed in this application:

| Results from home phase of G170267 | Control IQ | SAP | F | p value |
|---|---|---|---|---|
| Percent between 70 and 180mg/dl | $71 \pm 6.6$ | $52.8 \pm 13.5$ | 16.4 | 0.001 |

- 1430 From the DCLP1 study using the same algorithm in an older cohort, the effective standard
- deviation (after adjusting for the correlation between baseline and follow up) for time in range 70-
- 180 mg/dL over the course of 6 months was 6% (95% CI 5% to 7%) for the CLC group and 7%
- 1433 (95% CI 6% to 8%) for the SAP group.
- 1434 A total sample size was computed to be N=60 for the following assumptions: (1) 3:1 [CLC:SC]
- randomization, (2) 90% power, (3) a 10% absolute increase in % time in range 70-180 mg/dL, (4)
- an effective SD of 10%, and (5) 2-sided type 1 error of 0.05.

- 1437 The total sample size has been increased to N=100 to account for dropouts and to increase the
- number of participants who will be exposed to the CLC system for an enhanced safety and
- 1439 feasibility assessment.
- 1440 11.4 Efficacy Outcome Measures
- 1441 11.4.1 Primary Efficacy Endpoint
- CGM-measured % in range 70-180 mg/dL
- 1443 11.4.2 Secondary Efficacy Endpoints
- 1444 11.4.2.1 Secondary Efficacy Endpoints Included in Hierarchical Analysis
- 1445 The following secondary endpoints will be tested in a hierarchical fashion as described in
- 1446 section 11.7.1.
- CGM-measured % above 180 mg/dL
- CGM-measured mean glucose
- HbA1c at 16 weeks
- CGM-measured % below 70 mg/dL
- CGM-measured % below 54 mg/dL
- CGM-measured % above 250 mg/dL
- Glucose variability measured with the coefficient of variation (CV)
- 1454 11.4.2.2 Other Secondary Efficacy Endpoints
- 1455 The following endpoints are considered exploratory. Type 1 error for these endpoints will be
- 1456 controlled using the false discovery rate (FDR) instead of the familywise error rate (FWER).
- 1457 *CGM-Measured*:
- 1458 % in range 70-140 mg/dL
- glucose variability measured with the standard deviation (SD)
- 1460 % <60 mg/dL
- low blood glucose index
- hypoglycemia events (defined as at least 15 consecutive minutes <70 mg/dL)
- 1463 % > 300 mg/dL
- high blood glucose index
- % in range 70-180 mg/dL improvement from baseline to 16 weeks ≥5%
- % in range 70-180 mg/dL improvement from baseline to 16 weeks ≥10%

#### 1467 *HbA1c*:

- 1468 HbA1c < 7.0% at 16 weeks
- HbA1c <7.5% at 16 weeks
- HbA1c improvement from baseline to 16 weeks >0.5%
- HbA1c improvement from baseline to 16 weeks >1.0%
- HbA1c relative improvement from baseline to 16 weeks >10%
- HbA1c improvement from baseline to 16 weeks >1.0% or HbA1c <7.0% at 16 weeks

#### 1474 *Questionnaires*

- Fear of Hypoglycemia Survey (HFS-II) total score, 2 subscales and 4 factor scores:
- ◆ Behavior (avoidance and maintain high BG)
- ♦ Worry (helplessness and social consequences)
- Clarke Hypoglycemia Awareness Scores
- Problem Areas In Diabetes Survey (PAID)
- INSPIRE survey scores
- PedsQL Diabetes Module total score and 5 subscales:
- 1482 ♦ Diabetes
- 1483 ♦ Treatment I
- 1484 ♦ Treatment II
- 1485 ♦ Worry
- 1486 ♦ Communication
- Pittsburgh Sleep Quality Index (Parent only)
- System Usability Scale (SUS)
- 1489 *Other:*
- 1490 Insulin
- ↑ Total daily insulin (units/kg)
- 1492 ♦ Basal: bolus insulin ratio
- Weight and Body Mass Index (BMI)

#### 1494 11.4.3 CGM Metrics Calculations

- Randomization is preceded by two weeks of CGM run-in, which will be used in the calculation
- of baseline CGM metrics. For participants who are eligible to skip the run-in, comparable

| 1497<br>1498 | amount of CGM data from their own sensors will be taken before randomization visit to calculate baseline CGM metrics. |
|---|---|
| 1499<br>1500<br>1501 | CGM data starting from randomization visit through the 16-week visit will be included in the calculation of each CGM metric. Percentages in range 70-180 mg/dL (and all other CGM-based metrics) will be calculated giving equal weight to each CGM point for each participant. |
| 1502 | 11.5 Analysis Datasets and Sensitivity Analyses |
| 1503<br>1504<br>1505 | All analyses comparing the CLC arm with SC arm will follow the intention-to-treat (ITT) principle with each participant analyzed according to the treatment assigned by randomization. All randomized participants will be included in the primary and secondary hierarchical analyses. |
| 1506<br>1507 | Safety outcomes will be reported for all enrolled participants, irrespective of whether the participants was randomized or the study was completed. |
| 1508 | 11.5.1 Per Protocol Analyses |
| 1509<br>1510 | Per-protocol analyses will be performed for primary outcome and secondary hierarchical outcomes only if >5% of participants will be excluded: |
| 1511 | • CLC arm: Closed loop mode active for at least 80% of the time |
| 1512 | • SC arm: CGM use for at least 80% of the time |
| 1513 | 11.5.2 Other Sensitivity Analyses |
| 1514 | <u>Confounding</u> |
| 1515<br>1516<br>1517<br>1518<br>1519 | The primary analysis described below will include a pre-specified list of covariates. As an additional sensitivity analysis, any baseline demographic or clinical characteristics observed to be imbalanced between treatment groups will be added as covariates to the analyses of the primary endpoint. The determination of a meaningful baseline imbalance will be based on clinical judgement and not a p-value. |
| 1520 | Exclude First 2 Weeks of CGM Data |
| 1521<br>1522<br>1523<br>1524 | As noted above in Section 11.4.3, calculation of CGM metrics will include all available post-randomization CGM data. As a sensitivity analysis, CGM metrics will be recalculated by excluding the first two weeks of CGM data following the randomization visit. The primary analysis will be replicated based on the recalculated outcome. |
| 1525 | Missing Data |
| 1526<br>1527<br>1528 | It is worth emphasizing that any statistical method for handling missing data makes a number of untestable assumptions. The goal will be to minimize the amount of missing data in this study so that results and conclusions will not be sensitive to which statistical method is used. To that end, |

- sensitivity analyses will be performed to explore whether results are similar for primary analysis
- when using different methods. The following methods will be applied:
- Direct likelihood (primary analysis described below)
- Rubin's multiple imputation
- Multiple imputation with pattern mixture model
- Available cases only

### 1535 11.6 Analysis of the Primary Efficacy Endpoint

- Summary statistics (mean  $\pm$  SD or median (quartiles)) will be reported for the CGM-measured %
- in range 70-180 mg/dL and for differences from pre-randomization by treatment group.
- 1538 Changes from run-in pre-randomization CGM wear to the 16-week post-randomization period in
- 1539 CGM-measured % in range 70-180 mg/dL between two treatment arms will be compared using a
- linear mixed effects regression model while adjusting for baseline CGM-measured % in range
- 70-180 mg/dL, age, prior CGM and pump use, and clinical center (random effect). Missing data
- will be handled using direct likelihood. Residual values will be examined for an approximate
- normal distribution. If residuals are highly skewed, then a transformation or robust statistical
- method (e.g., non-parametric or MM estimation) will be used instead. It is expected that the
- residual values for CGM-measured % in range 70-180 mg/dL will follow an approximate normal
- 1546 distribution.

## 1547 11.7 Analysis of the Secondary Endpoints

- Point estimated and confidence intervals for the treatment arm differences will be presented for
- all secondary metrics. The models will adjust for the corresponding baseline metric, age, prior
- 1550 CGM and pump use, and clinical center (random effect).

#### 1551 11.7.1 Hierarchical Analyses

- To preserve the overall type 1 error for selected key secondary endpoints, a hierarchical testing
- procedure will be used. If the primary analysis for time in range described above results in a
- statistically significant result (p < 0.05), then testing (similar with the model described above
- for the primary outcome) will proceed to the next outcome metric in the following order:
- CGM-measured % in range 70-180 mg/dL (primary outcome)
- CGM-measured % above 180 mg/dL
- CGM-measured mean glucose
- 1559 HbA1c at 16 weeks
- CGM-measured % below 70 mg/dL
- CGM-measured % below 54 mg/dL
- CGM-measured % above 250 mg/dL

• Glucose variability measured with the coefficient of variation (CV)

This process continues iteratively moving to the next variable down on the list until a non-significant result ( $p \ge 0.05$ ) is observed, or all eight variables have been tested. If a non-significant result is encountered, then formal statistical hypothesis testing is terminated and any variables below on the list are not formally tested.

For example, in the hypothetical scenario depicted in the table below, the first four outcome variables all have a significant result so testing continues to the fifth variable (CGM % below 70 mg/dL). The result is not significant for that fifth variable (p = 0.06) so testing stops. No formal hypothesis test is conducted for the last three variables on the list in this example scenario.

| HIERARCHICAL<br>ORDER | OUTCOME<br>VARIABLE | TREATMENT<br>ARM P-VALUE | SIGNIFICANT? | ACTION |
|---|---|---|---|---|
| 1 <sup>st</sup> | CGM % 70-180 mg/dL (primary outcome) | 0.001 | Yes | Test next variable |
| $2^{\mathrm{nd}}$ | CGM % above 180 mg/dL | 0.02 | Yes | Test next variable |
| 3 <sup>rd</sup> | CGM mean glucose | 0.007 | Yes | Test next variable |
| 4 <sup>th</sup> | HbA1c at 16 weeks | 0.03 | Yes | Test next variable |
| 5 <sup>th</sup> | CGM % below 70 mg/dL | 0.06 | No | Stop formal testing |
| 6 <sup>th</sup> | CGM % below 54 mg/dL | Not tested | Unknown | N/A |
| 7 <sup>th</sup> | CGM % above 250 mg/dL | Not tested | Unknown | N/A |
| 8 <sup>th</sup> | Glucose CV | Not tested | Unknown | N/A |

### **Table 6. Example Hypothetical Hierarchical Test Results**

- Regardless of the results of the hierarchical testing, summary statistics appropriate to the
- distribution will be tabulated by treatment arm for each hierarchical outcome. A 95% confidence
- 1575 interval for the treatment arm difference will also be calculated for all seven secondary
- 1576 hierarchical outcomes listed above. However, a confidence interval that excludes zero will not
- be considered a statistically significant result if an outcome variable higher on the hierarchical
- list failed to reach statistical significance.

#### 11.7.2 Other Endpoint Analyses

# 1580 <u>CGM-Measured Outcomes</u>

- The analyses for the secondary CGM-measured outcomes will parallel those mentioned above
- for the primary outcome. For the binary CGM outcomes, risk-adjusted percentages by treatment
- group will be calculated from a logistic regression model.

#### 1584 *HbA1c*

1564

1565

1566 1567

1568 1569

1570

1571

1572

1579

- Summary statistics (mean  $\pm$  SD) will be reported for the central lab HbA1c at baseline, 16 weeks
- and for differences from pre-randomization by treatment group.

- 1587 Change in HbA1c from baseline to 16 weeks will be compared between the two treatment arms
- using a linear model while adjusting for baseline HbA1c, age, prior CGM and pump use, and
- 1589 clinical center (random factor).
- 1590 For extension phase, efficacy of the AP will be compared by using the final 12 weeks of the
- 1591 control period vs. the 12-week AP extension phase. Each participant will be their own control.
- 1592 Missing data will be handled using direct likelihood in a regression model including all available
- 1593 central laboratory HbA1c measurements at baseline and 16-week visits. When available, the
- local HbA1c measurement will be included in the regression model as an auxiliary variable.
- For the binary HbA1c outcomes listed above, risk-adjusted percentages by treatment group will
- be computed from a logistic regression model. The logistic regression will adjust for the same
- factors mentioned above for the analysis with HbA1c as a continuous factor (i.e., baseline
- 1598 HbA1c, age, prior CGM and pump use, and clinical center as a random effect).
- 1599 *Questionnaires and Other Outcomes*
- 1600 For questionnaires administered to both randomization groups, comparisons will be made using
- similar linear models as described above for the primary outcomes. Separate models will be run
- 1602 for the total score and each of the subscales listed above.
- Similarly, for insulin, weight and BMI metrics comparisons will be made using similar linear
- models as described above for the primary HbA1c analysis.
- 1605 11.8 Safety Analyses
- All randomized participants will be included in these analyses and all their post-randomization
- safety events will be reported.
- Safety analyses of the main study (randomized trial phase) will include events occurring on or
- after randomization until and including the 16-week visit or Day 126 from randomization,
- whichever occurs first. Safety analyses of the extension phase will include subsequent events
- until the last visit date or the last event date (whichever is later).
- Any pre-randomization adverse events will be tabulated separately and will include all
- participants even if never randomized.
- For the following outcomes, mean  $\pm$  SD or summary statistics appropriate to the distribution will
- be tabulated by treatment group and formal statistical comparisons (main study phase only) will
- be performed if there are enough events (at least 5 events combined between the two treatment
- 1617 groups):
- Number of SH events and SH event rate per 100 person-years
- Number of DKA events and DKA event rate per 100 person-years
- Any adverse event' rate per 100 person-years

- Number of calendar days with any ketone level ≥1.0 mmol/L
- CGM-measured hypoglycemic events (≥15 minutes with glucose concentration <54 mg/dL)
- CGM-measured hyperglycemic events (≥15 minutes with glucose concentration >300 mg/dL)

1625

- 1626 If enough events, the numbers of SH/DKA events will be compared between the two treatment
- arms during the main study phase using a robust Poisson regression. The regression will adjust
- 1628 for the participant-reported number of events prior to the start of the study and clinical center as
- random effect. The amount of follow up will be included as an offset covariate to compare the
- rates. Similar analyses will be done for comparing any adverse event and number of calendar
- days with ketone events between the two treatment groups, except that clinical center will be the
- only covariate to be adjusted in the model.
- 1633 For CGM-measured hypoglycemia/hyperglycemia events, event rates per week will be compared
- using similar linear mixed effects regression models as described above for the primary outcome.

1635

- 1636 For both the main study and extension phases, the following safety outcomes will be tabulated by
- treatment group without a formal statistical comparison:
- Other serious adverse events (SAE)
- BG-measured hypoglycemic events (days with at least one BG record <54 mg/dL)
- BG-measured hyperglycemic events (days with at least one BG record >350 mg/dL)
- Worsening of HbA1c from baseline to 16 weeks by >0.5%
- Investigational device related (intervention group only):
- 1643 Adverse device effects (ADE)
- o Serious adverse device events (SADE)
- 0 Unanticipated adverse device effects (UADE)

1646

- 1647 11.9 Intervention Adherence
- 1648 The following tabulations and analyses will be performed by treatment group to assess
- intervention adherence for the study:
- Sensor use –percent time of use, overall and by 4-weekly
- The daily frequency of downloaded BGM use overall and by 4-weekly
- For CLC arm only, the following will be tabulated to assess adherence:
- % time in different operational modes overall and by 4-weekly

- 1654 11.10 Adherence and Retention Analyses
- 1655 The following tabulations and analyses will be performed by treatment group to assess protocol
- adherence for the study:
- Number of protocol and procedural deviations per participant along with the number and percentage of participants with each number of deviations
- Number of protocol and procedural deviations by severity with brief descriptions listed
- Flow chart accounting for all participants at all scheduled visits and phone contacts post treatment initiation to assess visit and phone completion rates
- Number of and reasons for unscheduled visits and phone calls
- Number of participants who stopped treatment and reasons
- 1664 11.11 Baseline Descriptive Statistics
- Baseline demographic and clinical characteristics of the cohort of all randomized participants
- will be summarized in a table using summary statistics appropriate to the distribution of each
- variable. Descriptive statistics will be displayed by treatment group.
- 1668 Will include:
- 1669 Age
- 1670 HbA1c
- 1671 Gender
- Race/Ethnicity
- Family income, education, and/or insurance status
- Insulin method before enrollment (pump vs. MDI)
- CGM use before enrollment
- 1676 Diabetes duration
- BMI (height and weight)
- 1678 C-peptide
- Participant-reported number of SH and DKA 12 months prior to the start of the study
- 1680 **11.12 Device Issues**
- The following tabulations and analyses will be performed by treatment group to assess device
- 1682 issues:
- Device malfunctions requiring study team contact and other reported device issues

- Sensor performance metrics (difference, absolute relative difference, and International Organization for Standardization criteria) if applicable, by sensor version.
- Rate of different failure events and alarms per 24 hours recorded by the Control-IQ system overall and by month

# 1688 11.13 Planned Interim Analyses

- All above efficacy and safety analyses will be conducted after all subjects completed the primary
- study phase. No sample size re-estimation will be needed for the extension phase. The data may
- be used for PMA, with no interruption on the extension phase.
- In addition, the DSMB will review safety data at intervals, with no formal stopping rules other
- than the guidelines provided in the participant-level and study-level stopping criteria (as defined
- in Section 9.5 of the protocol).

# 1695 11.14 Subgroup Analyses

- In exploratory analyses, the primary outcome (time 70-180 mg/dL), % time <70 mg/dL and HbA1c
- at 16 weeks will be assessed separately in various subgroups and for continuous variables
- according to the baseline value as defined below. Tests for interaction with treatment group will
- be performed and further explored if an interaction will be found in the first place.
- 1700 Interpretation of subgroup analyses will depend on whether the overall analysis demonstrates a
- significant treatment group difference. In the absence of such an overall difference and if
- performed, subgroup analyses will be interpreted with caution. For continuous variables, results
- will be displayed in subgroups based on cutpoints although the analysis will utilize the variable as
- 1704 continuous, except for age which will be analyzed both as a continuous variable and in two age
- groups. If there is insufficient sample size in a given subgroup, the cutpoints for continuous
- measures may be adjusted per the observed distribution of values. Cutpoint selection for display
- purposes will be made masked to the outcome data.
- 1708 Baseline HbA1c
- Baseline CGM time spent <70 mg/dL
- Baseline CGM time spent >180 mg/dL
- Baseline CGM time 70-180 mg/dL
- Device use before the enrollment: pump/MDI, CGM/no CGM, and combinations of both
- 1713 Age
- 1714 Sex
- 1715 Race/ Ethnicity
- 1716 Clinical center
- BMI (Height and weight)
- Family income, education, and/or insurance status

- 1719 C-peptide level
- 1720 11.15 Multiple Comparison/Multiplicity
- 1721 Primary Analysis
- 1722 Since there will be a single comparison for the primary outcome (CGM-measured % 70-180
- 1723 mg/dL), no adjustment is needed.
- 1724 Secondary Hierarchical Analyses
- 1725 The hierarchical testing procedure described above in section 11.7.1 will be used to control the
- overall type 1 error for the primary outcome plus seven key secondary outcomes identified above.
- 1727 All Other Secondary Analyses
- For all above-mentioned secondary analyses, the false discovery rate will be controlled using the
- adaptive Benjamini-Hochberg procedure.
- 1730 11.16 Exploratory Analyses
- 1731 In addition to the analysis for the CGM-measured endpoints described earlier, separate analyses
- will be conducted for daytime and nighttime.
- 1733 The CGM-measured analyses will be replicated with only CGM data when the closed-loop was
- active for the CLC group. The CGM data for the SC group will be the same as mentioned above
- in the CGM Metrics Calculation section 11.4.3.

# **Chapter 12: Data Collection and Monitoring**

## 1737 **12.1** Case Report Forms and Device Data

1736

- 1738 The main study data are collected through a combination of electronic case report forms
- 1739 (CRFs) and electronic device data files obtained from the study software and individual hardware
- 1740 components. These electronic device files and electronic CRFs from the study website are
- 1741 considered the primary source documentation.
- When data are directly collected in electronic case report forms, this will be considered the source
- data. Each participating clinical center will maintain appropriate medical and research records for
- 1744 this trial, in compliance with ICH E6 and regulatory and institutional requirements for the
- 1745 protection of confidentiality of participants.

# 1746 12.2 Study Records Retention

- 1747 Study documents should be retained for a minimum of 2 years after the last approval of a marketing
- application in an ICH region and until there are no pending or contemplated marketing applications
- in an ICH region or until at least 2 years have elapsed since the formal discontinuation of clinical
- development of the investigational product. These documents should be retained for a longer
- period, however, if required by local regulations. No records will be destroyed without the written
- 1752 consent of the sponsor, if applicable. It is the responsibility of the sponsor to inform the
- investigator when these documents no longer need to be retained.

# 1754 **12.3 Quality Assurance and Monitoring**

- Designated personnel from the Coordinating Center will be responsible for maintaining quality
- assurance (QA) and quality control (QC) systems to ensure that the clinical portion of the trial is
- 1757 conducted and data are generated, documented and reported in compliance with the protocol, Good
- 1758 Clinical Practice (GCP) and the applicable regulatory requirements. Adverse events will be
- 1759 prioritized for monitoring.
- 1760 A risk-based monitoring (RBM) plan will be developed and revised as needed during the course
- of the study, consistent with the FDA "Guidance for Industry Oversight of Clinical Investigations
- 1762 A Risk-Based Approach to Monitoring" (August 2013). Study conduct and monitoring will
- 1763 conform with 21 Code of Federal Regulations (CFR) 812.
- The data of most importance for monitoring at the clinical center are participant eligibility and
- adverse events. Therefore, the RBM plan will focus on these areas. As much as possible, remote
- monitoring will be performed in real-time with on-site monitoring performed to evaluate the verity
- and completeness of the key clinical center data. Elements of the RBM may include:
- Qualification assessment, training, and certification for clinical centers and clinical center personnel
- Oversight of Institutional Review Board (IRB) coverage and informed consent procedures
- Central (remote) data monitoring: validation of data entry, data edits/audit trail, protocol

- review of entered data and edits, statistical monitoring, study closeout
- On-site monitoring (site visits): source data verification, site visit report
- Agent/Device accountability
- Communications with clinical center staff
- Participant retention and visit completion
- Quality control reports
- Management of noncompliance
- Documenting monitoring activities
- Adverse event reporting and monitoring
- 1781 Coordinating Center representatives or their designees may visit the study facilities at any time
- in order to maintain current and personal knowledge of the study through review of the records,
- 1783 comparison with source documents, observation and discussion of the conduct and progress of the
- 1784 study.
- 1785 **12.4 Protocol Deviations**
- 1786 A protocol deviation is any noncompliance with the clinical trial protocol, GCP, or procedure
- requirements. The noncompliance may be either on the part of the participant, the investigator, or
- the clinical center staff. As a result of deviations, corrective actions are to be developed by the
- 1789 clinical center and implemented promptly.
- 1790 The clinical center PI/study staff is responsible for knowing and adhering to the IRB requirements.
- 1791 Further details about the handling of protocol deviations will be included in the monitoring plan.

# Chapter 13: Ethics/Protection of Human Participants

#### 1793 13.1 Ethical Standard

1792

1797

1804

1805

- 1794 The investigator will ensure that this study is conducted in full conformity with Regulations for
- the Protection of Human Participants of Research codified in 45 CFR Part 46, 21 CFR Part 50, 21
- 1796 CFR Part 56, and/or the ICH E6.

#### 13.2 Institutional Review Boards

- 1798 The protocol, informed consent form(s), recruitment materials, and all participant materials will
- be submitted to the IRB for review and approval. Approval of both the protocol and the consent
- 1800 form must be obtained before any participant is enrolled. Any amendment to the protocol will
- require review and approval by the IRB before the changes are implemented to the study. All
- changes to the consent form will be IRB approved; a determination will be made regarding whether
- previously consented participants need to be re-consented.

#### 13.3 Informed Consent Process

#### 13.3.1 Consent Procedures and Documentation

- 1806 Informed consent is a process that is initiated prior to the individual's agreeing to participate in the
- study and continues throughout the individual's study participation. Extensive discussion of risks
- and possible benefits of participation will be provided to the participants and their families.
- 1809 Consent forms will be IRB-approved and the participant will be asked to read and review the
- document. The investigator will explain the research study to the participant and answer any
- questions that may arise. All participants will receive a verbal explanation in terms suited to their
- comprehension of the purposes, procedures, and potential risks of the study and of their rights as
- research participants. Participants will have the opportunity to carefully review the written consent
- 1814 form and ask questions prior to signing.
- The participants should have the opportunity to discuss the study with their surrogates or think
- about it prior to agreeing to participate. The participant will sign the informed consent and child
- assent documents prior to any procedures being done specifically for the study. The participants
- 1818 may withdraw consent at any time throughout the course of the trial. A copy of the informed
- 1819 consent and child assent documents will be given to the participants for their records. The rights
- and welfare of the participants will be protected by emphasizing to them that the quality of their
- medical care will not be adversely affected if they decline to participate in this study.

# 1822 13.3.2 Participant and Data Confidentiality

- 1823 The study monitor, other authorized representatives of the sponsor, representatives of the IRB or
- device company supplying study product may inspect all documents and records required to be
- maintained by the investigator, including but not limited to, medical records (office, clinic, or
- hospital) for the participants in this study. The clinical center will permit access to such records.

- The study participant's contact information will be securely stored at each clinical center for internal use during the study. At the end of the study, all records will continue to be kept in a secure location for as long a period as dictated by local IRB and Institutional regulations.
- Study participant research data, which is for purposes of statistical analysis and scientific reporting, 1830 1831 will be transmitted to and stored at the Jaeb Center for Health Research and the University of Virginia Center for Diabetes Technology. This will not include the participant's contact or 1832 identifying information. Rather, individual participants and their research data will be identified 1833 by a unique study identification number. The study data entry and study management systems 1834 used by clinical centers and by Jaeb research staff will be secured and password protected. At the 1835 1836 end of the study, all study databases will be de-identified and archived at Jaeb Center for Health Research and the University of Virginia Center for Diabetes Technology. Permission to transmit 1837
- data will be included in the informed consent.

- 1. Kovatchev, B.P., Breton, M.D., Keith-Hynes, P.T., Patek, S.D. The Diabetes Assistant (DiAs)

   Unified platform for monitoring and control of blood glucose levels in diabetic patients;

  PCT/US12/43910, 2012.
- Keith Hynes, P., Guerlain, S., Mize, L.B., Hughes Karvetski, C., Khan, M., McElwee Malloy,
   M. & Kovatchev, B.P. DiAs user interface: A patient-centric interface for mobile artificial
   pancreas systems. J Diabetes Sci Technol, 7, 1416–1426 (2013). PMID: 24351168
- Place, J., Robert, A., Ben Brahim, N., Keith Hynes, P., Farret, A., Pelletier, M.J., Buckingham,
   B., Breton, M., Kovatchev, B.P. & Renard, E. DiAs web monitoring: A real-time remote
   monitoring system designed for artificial pancreas outpatient trials. J Diabetes Sci Technol, 7,
   1427–1435. (2013). PMID: 24351169
- 4. Keith-Hynes, P., Mize, B., Robert, A., Place, J. The Diabetes Assistant: A smartphone-based system for real-time control of blood glucose. Electronics 2014, 3, 609-623; doi:10.3390/electronics3040609
- Kovatchev, B.P., Renard, E., Cobelli, C., Zisser, H., Keith-Hynes, P., Anderson, S.M. Brown,
   S.A. Chernavvsky, D.R., Breton, M.D., Farret, A., Pelletier, M.J., Place, J., Bruttomesso, D.,
   Del Favero, S., Visentin, R., Filippi, A., Scotton, R., Avogaro, A. & Doyle III, F.J. Feasibility
   of outpatient fully integrated closed-loop control: First studies of wearable artificial pancreas.
   Diabetes Care, 36, 1851-1858 doi: 10.2337/dc12-1965 (2013). PMID: 23801798, PMCID:
   PMC3687268
- Kovatchev, B.P., Renard, E., Cobelli, C., Zisser, H., Keith-Hynes, P., Anderson, S.M., Brown,
   S.A., Chernavvsky, D.R., Breton, M.D., Mize, L.B., Farret, A., Place, J., Bruttomesso, D., Del
   Favero, S., Boscari, F., Galasso, S., Avogaro, A., Magni, L., Di Palma, F., Toffanin, C.,
   Messori, M., Dassay, E., Doyle, F. III. Safety of outpatient closed-loop control: First
   randomized crossover trials of a wearable artificial pancreas. Diabetes Care, 37, 1789-1796
   doi: 10.2337/dc13-2076 (2014). PMID: 24929429, PMCID: PMC4067397
- 7. DeSalvo, D., Keith-Hynes, P., Peyser, T., Place, J., Caswell, K., Wilson, D., Harris, B., Clinton, P., Kovatchev, B.P., Buckingham, B.A. Remote glucose monitoring in camp setting reduces the risk of prolonged nocturnal hypoglycemia. Diabetes Technol Ther, 16, 1-7 doi:10.1089/dia.2013.0139 (2013). PMID: 24168317
- 8. Ly, T.T., Breton, M.D., Keith-Hynes, P., De Salvo, D., Clinton, P., Benassi, K., Mize, L.B., Chernavvsky, D.R., Place, J., Wilson, D.M., Kovatchev, B.P., Buckingham, B.A. Overnight glucose control with an automated, unified safety system in children and adolescents with type 1 diabetes at diabetes camp. Diabetes Care, 37, doi: 10.2337/dc14-0147 (2014). PMID: 24879841, PMCID: PMC4179507
- 9. Kropff, J., Del Favero, S., Place, J., Toffanin, C., Visentin, R., Monaro, M., Messori, M., Di Palma, F., Lanzola, G., Farret, A., Boscari, F., Galasso, S., Magni, P., Avogaro, A., Keith-Hynes, P., Kovatchev, B.P., Bruttomesso, D., Cobelli, C., DeVries, J.H., Renard, E., Magni, L., for the AP@home consortium. 2 month evening and night closed-loop glucose
- 1877 Magni, L., for the Ar@nome consortium. 2 month evening and fight closed-loop glucose control in patients with Type 1 Diabetes under free-living conditions: A randomised crossover

- trial. Lancet Diabetes Endocrinol, 3(12):939-47 dx.doi.org/10.1016/S2213-8587(15)00335-6 (2015).
- 1881 10. Renard, E et al. Reduction of hyper- and hypoglycemia during two months with a wearable artificial pancreas from dinner to breakfast in patients with type 1 diabetes. 2015-A-3083-
- Diabetes. American Diabetes Association 75th Scientific Sessions, Boston, MA, poster 940-P.
- 11. Anderson, S et al. First New Year's Night on closed-loop control (CLC) at home: Case reports from a multi-center international trial of long-term 24/7 CLC. 2015-A-4763-Diabetes. American Diabetes Association 75th Scientific Sessions, Boston, MA, presentation 223–OR.
- 12. Kovatchev BP. JDRF Multi-Center 6-Month Trial of 24/7 Closed-Loop Control. Advanced Technologies and Treatments for Diabetes (ATTD), Plenary Session, Milan, Italy, 2016.
- 13. Kovatchev, B.P. Closed-loop control modalities in type 1 diabetes: Efficacy and system acceptance. Advanced Technologies and Treatments for Diabetes (ATTD), Paris, France, 2015.
- 14. Del Favero S. A multicenter randomized cross-over Italian pediatric summer camp: AP vs SAP
   in 5-8 year old children. Advanced Technologies and Treatments for Diabetes (ATTD),
   Plenary Session, Milan, Italy, 2016.
- 1895 15. Cherñavvsky, D. et al. Closed-loop control during extended winter-sport exercise in youth with T1DM: Results from the first AP ski camp. ATTD Data Club Session, Milan, (2016).
- 16. Chernavvsky, D.R., DeBoer, M.D., Keith-Hynes, P., Mize, B., McElwee, M., Demartini, S., Dunsmore, S.F., Wakeman, C., Kovatchev, B.P., Breton, M.D. Use of an artificial pancreas among adolescents for a missed snack bolus and an underestimated meal bolus. Pediatric Diabetes, doi:10.1111/pedi.12230 (2014). PMID: 25348683
- 17. Brown, S.A., Kovatchev, B.P., Breton, M.D., Anderson, S.M., Keith-Hynes, P., Patek, S.D., Jiang, B., Ben Brahim, N., Vereshchetin, P., Bruttomesso, D., Avogaro, A., Del Favero, S., Boscari, F., Galasso, S., Visentin, R., Monaro, M., Cobelli, C. Multinight "bedside" closed-loop control for patients with type 1 diabetes. Diabetes Technol Ther 17(3), doi:10.1089/dia.2014.0259 (2015). PMID: 25594434, PMCID: PMC4346235
- 18. Kovatchev BP, Tamborlane WV, Cefalu WT, Cobelli C. The Artificial Pancreas in 2016: A Digital Treatment Ecosystem for Diabetes. Diabetes Care 2016; 39:1123-27. PMID: 27330124
- 19. Del Favero S, Boscari F, Messori M, Rabbone I, Bonfanti R, Sabbion A, IaFusco D, Schiaffini R, Visentin R, Calore R, Moncada YL, Galasso S, Galderisi A, Vallone V, Di Palma F, Losiouk E1, Lanzola G1, Tinti D, Rigamonti A, Marigliano M, Zanfardino A, Rapini N, Avogaro A,
- 1912 Chernavvsky D, Magni L, Cobelli C, Bruttomesso D. Randomized Summer Camp Crossover
- Trial in 5- to 9-Year-Old Children: Outpatient Wearable Artificial Pancreas Is Feasible and
- 1914 Safe. Diabetes Care. 2016;39:1180-5. PMID: 27208335
- 20. Renard E, Farret A, Kropff J, Bruttomesso D, Messori M, Place J, Visentin R, Calore R, Toffanin C, Di Palma F, Lanzola G, Galasso S, Avogaro A, Keith-Hynes P, Kovatchev BP,
- 1917 Del Favero S., Cobelli C, Magni L, DeVries HJ. AP@home Consortium. Day and night closed
- loop glucose control in patients with type 1 diabetes under free-living conditions: comparison

- of a single-arm, 1-month experience to results of a previously reported feasibility study of evening and night at home. Diabetes Care 2016; 39:1151-60. PMID: 27208331
- 1921 21. Anderson SM, Raghinaru D, Pinsker JE, Boscari F, Renard E, Buckingham BA, Nimri R,
- Doyle FJ III, Brown SA, Keith-Hynes P, Breton MD, Chernavvsky D, Bevier WC, Bradley
- 1923 PK, Bruttomesso D, Del Favero S, Calore R, Cobelli C, Avogaro A, Farret A, Place J, Ly TT,
- Shanmugham S, Phillip M, Dassau E, Dasanayake IS, Kollman C, Lum JW, Beck RW, and
- 1925 Kovatchev BP. Multinational home use of closed-loop control is safe and effective.
- 1926 Diabetes Care 2016; 39:1143-1150. PMID: 27208316
- 1927 22. DeBoer MD, Cherñavvsky DR, Topchyan K, Kovatchev BP, Francis GL, Breton MD. Heart
- rate informed artificial pancreas system enhances glycemic control during exercise in
- adolescents with T1D. Pediatr Diabetes. 2016; doi: 10.1111/pedi.12454. PMID: 27734563
- 1930 23. Kovatchev BP, Cheng P, Anderson SM, Pinsker JE, Boscari F, Buckingham BA, Doyle FJ.
- 1931 III, Hood KK, Brown SA. Breton MD, Chernavvsky DR, Bevier WC, Bradley PK,
- Bruttomesso D, Del Favero S, Calore R, Cobelli C, Avogaro A, Ly TT, Shanmugham S,
- Dassau E, Kollman C, Lum JW, Beck RW, for the Control to Range Study Group. Feasibility
- of Long-Term Closed-Loop Control: A Multicenter 6-Month Trial of 24/7 Automated Insulin
- 1935 Delivery. Diabetes Technol Ther 2017; 19: 18-24. doi:10.1089/dia.2016.0333. PMID:
- 1936 27982707
- 1937 24. DeBoer MD, Breton MD, Wakeman CA, Schertz EM, Emory EG, Robic JL, Kollar LL,
- 1938 Kovatchev BP, Chernavvsky DR. Performance of an Artificial Pancreas System for Young
- 1939 Children with Type 1 Diabetes. Diabetes Technol Ther 2017; 19, DOI: 10.1089/dia.2016.0424.
- 1940 PMID: 28426239
- 1941 25. Breton MD, Cherñavvsky DR, Forlenza GP, DeBoer MD, Robic J, Wadwa RP, Messer LH,
- Kovatchev BP, Maahs DM. Closed Loop Control During Intense Prolonged Outdoor Exercise
- in Adolescents With Type 1 Diabetes: The Artificial Pancreas Ski Study. Diabetes Care 2017
- 1944 Aug; dc170883. https://doi.org/10.2337/dc17-0883
- 1945 26. Ly TT, Gallego PH, Davis EA, Jones TW: Impaired Awareness of Hypoglycemia in a
- 1946 Population-Based Sample of Children and Adolescents With Type 1 Diabetes. Diabetes Care
- 1947 32(10):1802-1806, 2009
- 1948 27. Shepard JA, Vajda KA, Nyer M, Clarke WL, Gonder-Frederick LA, : Understanding the
- 1949 Construct of Fear of Hypoglycemia in Pediatric Type 1 Diabetes. J Pediatr Psychol 39(10):
- 1950 1115-1125, 2014
- 1951 28. Markowitz JT, Volkening LK, Butler DA, Antisdel-Lomaglio J, Anderson BJ, Laffel LM. Re-
- examining a measure of diabetes-related burden in parents of young people with Type 1
- diabetes: the Problem Areas in Diabetes Survey Parent Revised version (PAID-PR). Diabet
- 1954 Med. 2012;29(4):526–530. doi:10.1111/j.1464-5491.2011.03434.
- 1955 29. Varni, J. W., Delamater, A.M., Hood, K.K., Raymond, J.K., Chang, N.T., Driscoll, K.A.,
- Wong, J.C., Yi-Frazier, J.P., Grishman, E.K., Faith, M.A., Corathers, S.D., Kichler, J.C.,
- Miller, J.L., Doskey, E.M., Aguirre, V.P., Heffer, R.W., & Wilson, D. P. (in press). Pediatric
- 1958 Quality of Life Inventory (PedsQL) 3.2 Diabetes Module for youth with Type 2 diabetes:
- 1959 Reliability and validity. Diabetic Medicine.

- 30. J. Weissberg-Benchell, J.B. Shapiro, K. Hood, L.M. Laffel, D. Naranjo, K. Miller, K. Bernard:
   Assessing patient-reported outcomes for automated insulin delivery systems: the psychometric
   properties of the INSPIRE measures. *Diabet. Med.* 00: 1–9 (2019)
- 31. <u>Buysse DJ¹</u>, <u>Reynolds CF 3rd</u>, <u>Monk TH</u>, <u>Berman SR</u>, <u>Kupfer DJ</u>: The Pittsburgh Sleep
   Quality Index: a new instrument for psychiatric practice and research. <u>Psychiatry Res.</u> 1989
   May;28(2):193-213
- 32. Brown S, Raghinaru D, Emory E, Kovatchev B: First Look at Control-IQ: A New-Generation
   Automated Insulin Delivery System. Diabetes Care Oct 2018, dc181249; DOI: 10.2337/dc18 1249. PMID: 30305346
- 33. Ekhlaspour L, Wadwa RP, Chernavvsky D, Forlenza GP, Messer L, Town M, Swanson V,
   Maahs DM, Kovatchev B, Buckingham B, Breton M: Artificial Pancreas (AP) Ski Camp 2018:
   Successful Use of the Tandem Control-IQ AP System in Adolescents and Children During
   Winter Sports and at Home (abstract). Pediatric Diabetes 2018;17